Symphogen A/S Sym013-01

| P | Δ | R | F | X | $\mathbf{E}\mathbf{I}$ | . 1 | n | tei | rn | at | in | na | ı |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <b>┌</b> ┓ | | עוד | $\Delta$ | L' - | 1 | | | | 41 | .,, | 114 | |

Symphogen A/S

Sym013-01

An Open-label, Multicenter, Phase 1a/2a Trial Investigating the Safety, Tolerability and Antitumor Activity of Multiple Doses of Sym013 (Pan-HER), a Monoclonal Antibody Mixture Targeting EGFR, HER2 and HER3, in Patients with Advanced Epithelial Malignancies

**Statistical Analysis Plan** 

**Version: Final 1.0** 

**PAREXEL Project Number: 223277** 

# Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

#### **TABLE OF CONTENTS**

| 1 | INTRODUCTION | 11 |
|---|---|---|
| 2 | STUDY OBJECTIVES | |
| 2.1 | Objectives of Part 1, Dose-Escalation | |
| 2.1.1 | Primary Objective (Part 1) | |
| 2.1.2 | Secondary Objectives (Part 1) | |
| 3 | INVESTIGATIONAL PLAN | |
| 3.1 | Overall Study Design and Plan | |
| 3.2 | Endpoints and Associated Variables | 19 |
| 3.2.1 | Efficacy Variables | |
| 3.2.1. | 1 Tumor Response according to RECIST v1.1 | 20 |
| 3.2.1. | | |
| 3.2.2 | Pharmacodynamic, Biomarkers and Immunogenicity | 26 |
| 3.2.3 | Pharmacokinetic Variables | 27 |
| 3.2.4 | J | |
| 3.2.4. | 1 Dose Limiting Toxicity | 31 |
| 3.2.4. | | |
| 3.2.4. | 3 Clinical Laboratory and Pregnancy Test | 36 |
| 3.2.4. | 8 | |
| 3.2.4. | | |
| 3.2.4. | | |
| 3.2.4. | | |
| 3.2.4. | 8 Eastern Cooperative Oncology Group (ECOG) performance Status (PS) score | |
| 4 | STATISTICAL METHODS | |
| 4.1 | Data Quality Assurance | |
| 4.2 | General Presentation Considerations | 39 |
| 4.3 | Software43 | |
| 4.4 | Study Patients | |
| 4.4.1 | Disposition of Patients | |
| 4.4.2 | Protocol Deviations | |
| 4.5 | Analysis Sets | |
| 4.6 | Demographics and Baseline Characteristics, Disease History and Prior Cancer Therap | ies |
| | 44 | |
| | Medical History and Concomitant Illnesses | |
| 4.8 | Prior and Concomitant Medications | |
| 4.9 | Treatment Exposure and Compliance | |
| | Efficacy Evaluation | |
| 4.10. | | |
| | 1.1 Multi-center Studies | |
| | 1.2 Adjustments for Covariates | |
| | 1.3 Handling of Dropouts or Missing Data | |
| | eneral rules about handling of missing data refer to section 4.2. | |
| | 1.4 Multiple Comparisons/Multiplicity | |
| 4.10. | 1.5 Interim Analyses | 50 |

# Statistical Analysis Plan Template for Early Phase Studies

| Sympho | ogen A/S |
|--------|----------|
| Sym013 | 3-01 |

| 4.10. | 1.6 Examination of Subgroups50 | |
|---|---|---|
| 4.10.2 | 2 Analysis of Efficacy Variable(s) | |
| 4.10.2 | 2.1 Anti-Tumor Response according to RECIST v1.150 | |
| 4.10.2 | 2.2 Tumor Markers51 | |
| 4.10.3 | Pharmacodynamic, Biomarkers and Immunogenicity51 | |
| 4.10.3 | 3.1 Pharmacodynamic, Biomarkers, Immunogenicity (ADA) and Archival Tumor51 | |
| | 3.2 Skin Biopsy52 | |
| 4.10.3 | 3.3 Tumor Biopsy | |
| _ | Pharmacokinetics | |
| 4.10.4 | 4.1 Pharmacokinetic Concentrations | |
| 4.10.4 | 4.2 Handling of Values Below the Limit of Quantification (BLQ)56 | |
| 4.10.4 | 4.3 Pharmacokinetic Parameters | |
| 4.10.4 | 4.4 Pharmacokinetic Analysis56 | |
| 4.11 | Safety Evaluation | |
| 4.11. | The DLT Analysis Set will be used for evaluation of DLTs Dose Limiting Toxicities | |
| | (DLT)57 | |
| 4.11.2 | | |
| 4.11.3 | $\mathcal{E}$ | |
| 4.11.4 | Clinical Laboratory Evaluation60 | |
| 4.11.5 | 5 Electrocardiogram61 | |
| 4.11.6 | | |
| 4.11.7 | 7 Vital Signs and Body Measurements61 | |
| 4.11.8 | | |
| 4.11.9 | Eastern Cooperative of Oncology Group (ECOG) Performance Status (PS)62 | |
| 4.11. | | ıg |
| | Committee [DMC], Data and Safety Monitoring Board [DSMB])62 | |
| | Other Analyses62 | |
| | Determination of Sample Size62 | |
| 4.14 | Changes in the Conduct of the Study or Planned Analysis | |
| 5 | REFERENCES64 | |
| 6 | TABLES, FIGURES AND LISTINGS65 | |
| 7 | APPENDICES73 | |
| 7.1 | Schedule of Assessments Q1W dosing | |
| 7.2 | Schedule of Assessments Q2W dosing | |
| 7.3 | Derivation of CTCAE Grade – Hematological Tests | |
| 7.4 | Derivation of CTCAE Grade – Clinical Chemistry Tests | |
| 7.5 | Derivation of CTCAE Grade – Coagulation Tests | |

Symphogen A/S Sym013-01

### **REVISION HISTORY**

| Version No. | Effective Date | Summary of Change(s) |
|-------------|----------------|-----------------------------------------|
| Draft 0.1 | 28 Oct 2016 | New document |
| Draft 0.2 | May 2017 | Document Review |
| Draft 0.3 | 12 Feb 2019 | Document Review and Comments Resolution |
| Draft 0.4 | 07 March 2019 | Comments Resolution |
| Draft 0.5 | 27 March 2019 | Comments Resolution |
| Final 1.0 | 05 April 2019 | Final version for approval |

TP-GDO-WW-133-01 CONFIDENTIAL Project Document Version No. Final 1.0 Effective Date: 05 Sep 18 Project Document Effective Date: 05 April 2019 Related to: SOP-GDO-WW-019 

Symphogen A/S Sym013-01

#### LIST OF ABBREVIATIONS

List and define all acronyms and abbreviations used in the document here. Abbreviations should be spelled out in full and the abbreviation indicated in parentheses at first appearance in the text. Abbreviations should appear in alphabetical order.

| Abbreviation / Acronym | Definition / Expansion |
|---|---|
| 1M FUP | 1-Month Follow-up |
| ADA | Anti-Drug Antibody |
| ADC | Antibody Drug Conjugate |
| ADCC | Antibody-Dependent Cellular Cytotoxicity |
| AE | Adverse event |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| ANC | Absolute Neutrophil Count |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical therapeutic chemical |
| AUC | Area under the concentration-time curve |
| $AUC_{norm,\tau}$ | Dose normalized area under the concentration-time curve in a |
| | dosing interval, calculated as AUC $_{\mbox{\tiny T}}$ divided by the dose infused |
| $\mathrm{AUC}_{	au}$ | Area under the concentration-time curve in a dosing interval (i.e. |
| | from time zero (end of infusion) up to 168 hours). |
| $\mathrm{AUC}_{	au0}$ | Area under the concentration-time curve from start of infusion up |
| | to 168 hours. $AUC_{\tau 0}$ will be calculated similar to $AUC_{\tau}$ |
| BID | Bis in die (twice daily) |
| BLQ | Below the lower limit of quantification |
| BMI | Body Mass Index |
| BOR | Best Objective Response |
| BP | Blood pressure |
| Bpm | Beats per minute |


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 **Project Document Version No.** Final 1.0 **Project Document Effective Date**: 05 April 2019


Symphogen A/S Sym013-01

| Abbreviation / Acronym | Definition / Expansion |
|---|---|
| BUN | Blood Urea Nitrogen |
| C#/D# | Cycle #/ Day # |
| $C_{avg}$ | Average concentration at steady state |
| CDC | Complement-Dependent Cytotoxicity |
| $C_{EOI}$ | Concentration at End of Infusion |
| CI | Confidence interval |
| $CL_S$ | Clearance after first dose |
| $CL_{SS}$ | Clearance after 3 <sup>rd</sup> /4 <sup>th</sup> dose |
| $C_{max}$ | Maximum concentration |
| $C_{trough}$ | Trough concentration |
| CNS | Central Nervous System |
| CR | Complete Response |
| CRC | Colorectal Cancer |
| CRF | Case Report Form |
| CSP | Clinical Study Protocol |
| $C_{max}$ | Maximum observed concentration |
| $C_{\min}$ | Minimum observed concentration in the dosing interval |
| CS | Clinically significant |
| $C_{\mathrm{av,ss}}$ | Average concentration at steady state |
| $C_{max,ss}$ | Maximum observed concentration at steady state |
| $C_{\min,ss}$ | Minimum observed concentration at steady state |
| $C_{trough}$ | Concentration immediately prior to dosing |
| CT | Computed Tomography |
| CTCAE v4.03 | Common Terminology Criteria for Adverse Events (Version 4.03) |
| CTR | Clinical Trial Report |
| CV | Coefficient of variation |
| CYP | Cytochrome P450 |
| d | decimal places in the original reported value |
| DBP | Diastolic blood pressure |


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 Project Document Version No. Final 1.0 Project Document Effective Date: 05 April 2019 

Symphogen A/S Sym013-01

| Abbreviation / Acronym | Definition / Expansion |
|---|---|
| DCR | Disease Control Rate |
| CSR | Clinical Study Protocol |
| DLT | Dose-Limiting Toxicity |
| DMP | Data Management Plan |
| d.p. | decimal places |
| DSUR | Development Safety Update Report |
| DRM | Data Review Meeting |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| ЕСНО | Echocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| EGFR | Epidermal Growth Factor Receptor |
| EOI | End of Infusion |
| EOT | End-of-Treatment |
| FAS | Full Analysis Set |
| FDG | Fluorodeoxyglucose |
| GCP | Good Clinical Practice |
| GnRH | Gonadotropin-Releasing Hormone |
| НА | Health Authority |
| HER | Human Epidermal Growth Factor Receptor |
| HIV | Human Immunodeficiency Virus |
| HR | Heart rate |
| HRT | Hormone Replacement Therapy |
| IB | Investigator's Brochure |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation of Technical |
| | Requirements for Pharmaceuticals for Human Use |
| IgG1 | Immunoglobulin G1 |
| IHC | Immunohistochemistry |


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 Project Document Version No. Final 1.0 Project Document Effective Date: 05 April 2019 

Symphogen A/S Sym013-01

| Sym013-01 Abbreviation / Acronym | Definition / Expansion |
|---|---|
| IMP | Investigational Medicinal Product |
| INR | International Normalized Ratio |
| IRB | Institutional Review Board |
| IRR | Infusion-Related Reaction |
| IV | Intravenous |
| KRAS | Kirsten Rat Sarcoma Viral Oncogene Homolog |
| L | Linearity index |
| LLN | Lower Limit of Normal |
| LLOQ | Lower limit of quantification |
| LOQ | Limit of quantification |
| LVEF | Left Ventricular Ejection Fraction |
| mAb | Monoclonal Antibody |
| MAD | Maximum Administered Dose |
| MAPK | Mitogen-Activated Protein Kinase |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic Resonance Image/Imaging |
| mRNA | Messenger ribonucleic acid |
| MTD | Maximum tolerated dose |
| MUGA | Multi-Gated Acquisition |
| NA | Not available |
| NE | Not Evaluable |
| NCS | Not clinically significant |
| NK | Not known |
| NOAEL | No Observed Adverse Event Level |
| NRAS | Neuroblastoma RAS Viral Oncogene Homolog |
| NSAID | Nonsteroidal Anti-Inflammatory Drug |
| NSCLC | Non-Small Cell Lung Cancer |
| OR | Objective Response |
| OS | Overall Survival |


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 Project Document Version No. Final 1.0 Project Document Effective Date: 05 April 2019 

Symphogen A/S Sym013-01

| Abbreviation / Acronym | Definition / Expansion |
|---|---|
| OTC | Over the counter |
| PD | Pharmacodynamic or Progressive Disease (meaning to be |
| | extrapolated by the context) |
| PDs | Protocol Deviations |
| PET | Positron Emission Tomography |
| PI3K | Phosphoinositide 3-Kinase |
| PK | Pharmacokinetic |
| PO | Orally, by mouth |
| PR | Partial Response |
| PS | Performance Status |
| PSA | Prostate-Specific Antigen |
| PT | Prothrombin Time or Preferred Term (meaning to be extrapolated |
| | by the context) |
| PTT | Partial Thromboplastin Time |
| Q1W | Every week, weekly |
| Q2W | Every second week |
| QT | The QT interval is measured from the beginning of the QRS |
| | complex to the end of the T wave |
| QTc | corrected QT interval |
| QTcB | QT corrected using Bazzett's formula |
| QTcF | QT corrected using Fridericia's formula |
| RAS | Rat Sarcoma |
| RDI | Relative Dose Intensity |
| RECIST v1.1 | Response Evaluation Criteria in Solid Tumors (Version 1.1) |
| RP2D | Recommended Phase 2 Dose |
| RTK | Receptor Tyrosine Kinase |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic blood pressure |


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 Project Document Version No. Final 1.0
Project Document Effective Date: 05 April 2019


Symphogen A/S Sym013-01

| Abbreviation / Acronym | Definition / Expansion |
|---|---|
| SCCHN | Squamous Cell Carcinoma of the Head and Neck |
| SD | Standard Deviation or Stable Disease (meaning to be extrapolated |
| | by the context) |
| SE | Standard error of the mean |
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |
| SOI | Start of Infusion |
| SOP | Standard Operating Procedure(s) |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TBD | To Be Determined |
| TEAE | Treatment-emergent adverse event |
| TKI | Tyrosine Kinase Inhibitor |
| $t_{max}$ | Time to reach maximum concentration |
| TTP | Time To Progression |
| $T_{\frac{1}{2}}$ | Terminal elimination half-life |
| ULN | Upper Limit of Normal |
| $V_S$ | Volume of distribution during the terminal phase after first dose |
| $V_{SS}$ | Volume of distribution during the terminal phase after 3 <sup>rd</sup> /4 <sup>th</sup> dose |
| WHO-DD | World Health Organisation - Drug Dictionary |
| WT | Wild-Type |
| $\lambda_{ m z}$ | Terminal rate constant |


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

1 INTRODUCTION

The investigational medicinal product (IMP) tested in this trial is Sym013, referenced as Pan-

HER. Pan-HER is a recombinant antibody mixture containing 6 humanized immunoglobulin G1

(IgG1) mAbs, which bind specifically to non-overlapping epitopes on the EGFR (Hu1277 and

Hu1565), HER2 (Hu4384 and Hu4517) and HER3 (Hu5038 and Hu5082).

This is the first clinical trial to study Pan-HER.

HER family expression heterogeneity and plasticity in response to therapeutic intervention are

important drivers of primary and acquired drug resistance and pose challenges to effective cancer

treatment in the clinic. By targeting three receptors of the HER family, Pan-HER effectively

inhibits a range of cancers of various tissue origin and genetic background, including cell lines and

xenograft models with acquired resistance to therapeutic antibodies. Importantly, by down

modulating all three targets simultaneously, Pan-HER prevents compensatory receptor up-

regulation and renders the receptors unavailable for ligand binding and activation. Pan-HER

represents a novel strategy to deal with primary and acquired resistance and thus may provide a

clinically relevant effect in patient populations for which few therapeutic options exist.

Pan-HER is developed for the treatment of patients with resistant or refractory epithelial

malignancies. Initially, the safety and efficacy of Pan-HER are investigated in advanced epithelial

malignancies. Future development of Pan-HER may include pancreatic, esophageal, gastric, CRC,

NSCLC, advanced ovarian, and HER2-postive breast cancer having failed HER2 targeted therapy.

The Statistical Analysis Plan (SAP) details the statistical methodology to be used in analyzing

study data and outlines the statistical programming specifications, tables, figures, and listings. It

describes the variables and populations, anticipated data transformations and manipulations, and

other details of the analyses not provided in the clinical study protocol. This SAP covers the

planned analysis of all data collected on paper (source documents /case report forms [CRFs]),

captured electronically in DataLabs®, and provided by external vendors. PK/PD and

immunogenicity blood samples are analyzed by external laboratory Eurofins Pharma. Tissue

samples are analyzed by external laboratory Histogenex. Biomarkers blood samples are analyzed


by external laboratory Guardant Health.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

The analyses described are based on Clinical Study Protocol (CSP) Final 7.0 incorporating

Amendment No.6, dated 14/Jun/2018, Amendment No. 5, dated 23/Jan/2018, Amendment No. 4,

dated 04/May/2017, Amendment No. 3, dated 26/Apr/2017, Amendment No. 2, dated

14/Nov/2016, Amendment No. 1, dated 03/Oct/2016 and original CSP Version Final 1.0, dated

13/Jun/2016. The analyses described are based upon electronic Case Report Form (eCRF), version

10.0 dated 18/Oct/2018.

The SAP will be finalized prior to database lock and describes the statistical analysis as it is

foreseen when the study is being planned. If circumstances should arise during the study rendering

this analysis inappropriate, or if in the meantime improved methods of analysis should come to

light, different analyses may be performed. If this occurs, Symphogen will determine how the

revision impacts the study and how the SAP revision should be implemented. The details of the

revision will be documented and described in the clinical study report (CSR).

The study was designed to include a Part 1 (Dose-Escalation) followed by a Part 2 (Dose-

Expansion).

During Part 1, Symphogen decided to stop the SYM013-01 enrollment. Therefore, no patient is

enrolled in Part 2.

All protocol objectives planned data collection and analyses for Part 2 of the study will be omitted


hereafter in this SAP.

Related to: SOP-GDO-WW-019


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

2 STUDY OBJECTIVES

2.1 Objectives of Part 1, Dose-Escalation

2.1.1 Primary Objective (Part 1)

To assess the safety and tolerability of Pan-HER when administered either Q1W or Q2W by IV

infusion to separate dose-escalation cohorts of patients with advanced epithelial malignancies

without available therapeutic options.

2.1.2 Secondary Objectives (Part 1)

1. To determine a recommended phase 2 dose (RP2D) and regimen of Pan-HER

2. To evaluate the pharmacokinetic (PK) profile of Pan-HER

3. To evaluate the immunogenicity of Pan-HER

4. To evaluate target engagement in skin biopsy tissue (EGFR and HER3) and tumor biopsy tissue,

if available, (EGFR, HER2 and HER3)

5. To evaluate other potential pharmacodynamic biomarkers of Pan-HER action, and estimate, if

feasible, the magnitude of biological activity in peripheral blood and in skin biopsy (and tumor

biopsy, if available) tissue

6. To make a preliminary evaluation of the antitumor effect of Pan-HER

3 INVESTIGATIONAL PLAN

3.1 Overall Study Design and Plan

This is an open-label, multicenter trial composed of 2 parts in which Pan-HER will be evaluated

when administered by the IV route to patients with advanced epithelial malignancies without

available therapeutic options:

• Part 1 is a Phase 1a dose-escalation evaluating Q1W and Q2W schedules of administration

in separate dose-escalation cohorts to determine the RP2D and regimen of Pan-HER.


Related to: SOP-GDO-WW-019

#### Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

- During Part 1, cohorts of patients will receive increasing doses of Pan-HER on either Q1W or a Q2W schedule until establishment of the following for each schedule:
  - A maximum administered dose (MAD), the highest dose level administered (in mg/kg).
  - o A maximum tolerated dose (MTD), the highest dose of SYM013 with <33% patients who have experienced dose limiting toxicity (DLT) as defined by the protocol during cycle 1 of study treatment. Q1W and Q2W regimens may have different MTDs;
  - o A RP2D, determined based safety of Q1W and Q2W dose regimens as well as available PK and target engagement results, was to be identified. The RP2D may be equal to or lower than the MTD for the Q1W and/or Q2W dosing regimens.

The Part 1 starting dose of Pan-HER will be 1.0 mg/kg Q1W. The following dose levels of Pan-HER are planned to be evaluated:

#### Q1W

• Dose Level 1: 1 mg/kg Q1W

• Dose Level 2: 2 mg/kg Q1W

• Dose Level 3: 4 mg/kg Q1W

• \*Dose Level 4P: 6 mg/kg Q1W + P (lower doses with prophylaxis may be explored, if indicated)

• \*Dose Level 5P: 9 mg/kg Q1W + P

• \*Dose Level 6P: 12 mg/kg Q1W + P (no patient enrolled in this dose level)

• \*Dose Level 7P: 15 mg/kg Q1W + P (no patient enrolled in this dose level)


• \*Dose Level 8P: 18 mg/kg Q1W + P (highest potential dose allowed per protocol) (no patient

enrolled in this dose level)

**Project Document Effective Date**: 05 April 2019


Symphogen A/S Sym013-01

Q2W

• Dose Level 4: 6 mg/kg Q2W

• Dose Level 5: 9 mg/kg Q2W

• \*Dose Level 5P: 9 mg/kg Q2W+ P

• \*Dose Level 6P: 12 mg/kg Q2W+ P

• \*Dose Level 7P: 15 mg/kg Q2W + P

• \*Dose Level 8P: 18 mg/kg Q2W + P (highest potential dose allowed per protocol) (no patient

enrolled in this dose level)

\*Mandatory intensive IRR and oropharyngeal mucositis prophylaxis; 4-hour infusion (designated "P")

Note: Patients entered to Dose Levels 1, 2 and 3 were treated Q1W. As of Amendment 3, the dosing schedule in this trial was changed to Q2W. Patients entered to the trial prior to implementation of this amendment could continue to be treated Q1W.

Note: As of Amendment 5, patients entered to Dose Level 5P and all patients thereafter must receive intensive prophylaxis on a mandatory basis to reduce the risk of IRRs and oropharyngeal mucositis, and must receive Pan-HER over a fixed (at minimum) 4-hour (+10 min) period unless further prolongation is required for an individual patient due to the occurrence of an IRR. For patients entered to the trial prior to Amendment 5, these changes could be implemented at the Investigator's discretion based on the individual patient's prior experience with Pan-HER dosing.

Note: As of Amendment 6, Q1W dosing is reintroduced under the prophylaxis and infusion duration conditions outlined in Amendment 5. All patients must receive intensive prophylaxis, as defined herein, on a mandatory basis to reduce the risk of IRRs and oropharyngeal mucositis, and must receive Pan-HER infusions over a fixed (at minimum) 4-hour (+10 min) period, unless further prolongation is required for an individual patient due to the occurrence of an IRR. Reevaluation of Q1W dosing will begin at the 6 mg/kg dose; however, lower doses may be explored if indicated based on tolerability.

Initially, one patient will be treated at each dose level until the occurrence of a toxicity during Cycle 1 that activates the stopping rule of the single-patient cohort titration design. If such a toxicity has not occurred in the first 3 cohorts (i.e., cohorts of 1 mg/kg, 2 mg/kg, and 4 mg/kg


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

Q1W), the next cohort to open will be a 3-patient cohort and the design will switch to the 3+3

design.

Further dose-escalation will follow a standard 3+3 design with a target toxicity level of < 33% as

determined by the number of cycle 1 DLTs.

During Part 1, intermediate dose level(s) between 2 planned dose levels may be evaluated to further

characterize safety and tolerability of Pan-HER, if indicated based on toxicity observations and/or

results from PK and/or target engagement analyses.

A safety monitoring committee (SMC) will be established and will include Investigator(s),

Medical Monitor(s) and Sponsor's medical representatives. The SMC will review clinical and

laboratory safety data regularly throughout the trial and will select the RP2D and regimen to be

used in Part 2 based on safety data, as well as available PK and target engagement results.


The trial design is shown in Figure 1.

The overall Trial Plan is reported in Table - Overall Trial Plan.


Symphogen A/S Sym013-01

#### Figure 1 Overall Trial Design



Abbreviations: DLT: dose-limiting toxicity, G2T: grade 2 toxicity, M4D: maximum administered dose, MTD: maximum tolerated Dose; P(\*): prophylaxis; RP2D: recommended phase 2 dose; Q1W: every week; Q2W: every second week


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 Project Document Version No. Final 1.0 Project Document Effective Date: 05 April 2019 

Symphogen A/S Sym013-01

**Table - Overall Trial Plan** 

| <b>Screening Period</b> | |
|---|---|
| Screening | 14 days within first dose of Pan-HER |
| Treatment Period | |
| Treatment Allocation | The allocated dose and schedule of Pan-HER will depend upon cohort assignment and will be confirmed by Sponsor or designee on the <a href="Screening">Screening</a> and Allocation Form. |
| Pan-HER | Pan-HER will be initiated on C1/D1 and based on cohort assignment, will be administered either Q1W or Q2W to separate dose-escalation cohorts of patients by IV infusion in cycles of treatment: • Q1W: Dosing on Day 1, 8, 15, and 22 of each 28-day cycle (±2 days) • Q2W: Dosing on Day 1 and 15 of each 28-day cycle (±2 days) The duration of infusion will be (effective with Amendment 5): • Minimum of 4 hours (+10 min) for all infusions. Titrated rate increases during infusions, and infusion duration reductions after C1/D1, will no longer be allowed. For Part 1 of the trial, Pan-HER will be administered following delivery of intensive prophylaxis, as defined herein, on a mandatory basis to reduce the risk of IRRs and oropharyngeal mucositis. |
| Discontinuation of | Treatment will continue until unacceptable toxicity or other conditions |
| Pan-HER | preventing further treatment, PD, termination of the trial, or patient's decision to withdraw. |
| End of Treatment | |
| End of Treatment<br>Visit | Within 10 days after the decision to discontinue Pan-HER, an EOT Visit should be performed. |


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 Project Document Version No. Final 1.0
Project Document Effective Date: 05 April 2019


Symphogen A/S Sym013-01

| Follow-up | |
|---|---|
| One Month Follow- | Follow-up continues until 1 month (30+7 days) after the last dose of |
| up Visit | Pan-HER. At that time, a 1M FUP Visit should be performed. This visit constitutes the end of trial participation for the patient. |

Abbreviations (in alphabetical order): C1/D1, Cycle1/Day1; CR, complete response; EOT, End of Treatment Visit; IRR, infusion related reaction; IV, intravenous; 1M FUP, 1-Month Follow-up Visit; OS, overall survival; PD, progressive disease; PR, partial response; SD, stable disease.

#### 3.2 Endpoints and Associated Variables

Refer to the Schedule of Assessments for timing of assessments.

#### Primary Endpoint - Part 1, Dose-Escalation

The primary objective of the dose-escalation part is to assess the safety and tolerability of Pan-HER. This will be assessed by the primary endpoint for Part 1: occurrence of DLTs during Cycle 1 for each of the Pan-HER dose regimens.

#### **Secondary Efficacy Endpoints**

- Documented OR, defined as documented PR or CR, from baseline to end of trial participation (in patients with measurable disease only) (as measured in Part 1)
- Best overall response by RECIST v1.1, categorized as Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), and Not Evaluable (NE)
- Disease Control Rate (DCR)
- Changes in sum of diameters of target lesions from baseline to end of trial participation
- Time to documented PD (Time To Progression [TTP])

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

**Secondary Safety Endpoints** 

• Nature, incidence and severity of AEs measured from baseline to end of trial

participation

• AEs leading to dose-reductions, dose delays and permanent treatment cessation

Changes in safety laboratory values from baseline to end of trial participation

• Changes in vital signs and physical examinations from baseline to end of trial

participation

• Occurrence of ADA to Pan-HER measured in serum at selected timepoints from

baseline to end of trial participation

3.2.1 Efficacy Variables

3.2.1.1 Tumor Response according to RECIST v1.1

The anti-tumor activity of Pan-HER will be assessed according to RECIST, v 1.1 using CT or MRI.

The use of CT or MRI must be consistent per patient throughout the trial.

Disease Status Evaluation by CT or MRI will occur at:

Screening

Note: A CT/MRI performed within 28 days prior to Day 1 may be used for evaluation of

eligibility and as baseline scan, provided that the CT/MRI has been performed according

to the CTP requirements

• End of Cycle 2 and end of every second cycle thereafter, i.e. Cycle 4, 6, 8 etc.


Note: End of cycle assessments may be conducted at any time during the week prior to Day

1 of the next cycle

• After Suspected Progressive Disease (PD) (as soon as possible)

• Confirmation of response, to be performed 28 (+7) days after the first assessment of CR/PR

**Project Document Effective Date:** 05 April 2019


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

• EOT (if >3 weeks since previous CT/MRI)

• At 1M FUP (if PD was not documented before or at EOT)

If PD is documented at any time, no further disease assessments will be required. Patients with

documented PD will be discontinued from Pan-HER so that alternative management of their

malignancy may be considered.

For all imaging time points, the following will be recorded as per RECIST v1.1: Target lesions

including size, location, and type (nodal/non-nodal); sum of diameters of target lesions; any new

lesions noted during trial, including size, location, and type (nodal/non-nodal); response

assessment at each visit (PD, SD, PR, CR or Not Evaluable [NE]), per investigators evaluation.

Tumor evaluation according to RECIST 1.1 will be the basis for the derivation of all efficacy

endpoints. To be assigned a status of confirmed PR or CR, changes in disease status must be

confirmed by repeat imaging studies performed no less than 28 days (4 weeks) after the criteria

for response are first met. In the case of SD, follow-up measurements must have met the SD criteria

at least once after trial entry at a minimal interval in general no less than 6-8 weeks from first dose

of Pan-HER; for the scope of derivation of SD as best overall response, a minimal SD duration of

6 week will be required.

The following anti-tumor response endpoints will be derived based on Tumor evaluation according

to RECIST 1.1:

• Target and Non Target Response at each timepoint will be derived according to RECIST

1.1 [1].

o Evaluation of target lesions will be derived based on sum of diameters as

follow:

• 'Complete Response (CR): Disappearance of all target lesions. Any

pathological lymph nodes (whether target or non-target) must have

reduction in short axis to <10 mm.


Related to: SOP-GDO-WW-019

Symphogen A/S Sym013-01

■ Partial Response (PR): At least a 30% decrease in the sum of diameters

of target lesions, taking as reference the baseline sum diameters.

• Progressive Disease (PD): At least a 20% increase in the sum of

diameters of target lesions, taking as reference the smallest sum on

study (this includes the baseline sum if that is the smallest on study). In

addition to the relative increase of 20%, the sum must also demonstrate

an absolute increase of at least 5 mm. (Note: the appearance of one or

more new lesions is also considered progression).

• Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor

sufficient increase to qualify for PD, taking as reference the smallest

sum of diameters while on study.'

o Evaluation of non-target lesions: non-target lesions response will be reported in

CRF as CR, NON-CR/NON-PD, PD, Not Evaluated; worst response will be

taken as the Non-Target Lesion response for the correspondent timepoint; for

assessment of worst response the following order will be followed: PD, Not

Evaluated, NON-CR/NON-PD, CR.

Target and Non-Target Response at each timepoint, derived as described, will be reviewed

by Symphogen and PAREXEL on a patient by patient basis across time.

At each timepoint Overall Responses will be captured in CRF; as well Overall Responses

will also be derived according to RECIST 1.1 [1]:

Table 1 of above-mentioned paper [1] is reported below and will be used to derive overall

response at each time point for patients who have measurable disease at baseline. When

patients have non-measurable (therefore non-target) disease only, Table 2 is to be used.

Overall responses derived as described are supposed to coincide with overall responses

collected in CRF; cases of mismatch will be queried; any unsolved case of mismatch will

be reviewed by Symphogen and PAREXEL on a patient by patient basis across time.

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

**Project Document Effective Date**: 05 April 2019


Symphogen A/S Sym013-01

| Target lesions | Non-target lesions | New<br>lesions | Overall<br>response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or<br>not all evaluated | No | PR |
| SD | Non-PD or<br>not all evaluated | No | SD |
| Not all<br>evaluated | Non-PD | No | NE |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

| Non-target lesions | New lesions | Overall response |
|---|---|---|
| CR | No | CR |
| Non-CR/non-PD | No | Non-CR/non-PD |
| Not all evaluated | No | NE |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |
| CR = complete response NE = inevaluable. | e, PD = progressive | e disease, and |
| a 'Non-CR/non-PD' is pref | erred over 'stable dis | ease' for non-targe |

• Confirmed Best Overall Response (BOR) by RECIST v1.1.

#### Per RECIST 1.1[1]:

'the best overall response is the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation.' 'Specifically, in non-randomised trials where response is the primary endpoint, confirmation of PR or CR is needed to deem either one the 'best overall response'.' 'Best response determination in trials where confirmation of complete or partial response is

Symphogen A/S Sym013-01

required: Complete or partial responses may be claimed only if the criteria for each are met at a subsequent time point as specified in the protocol (generally 4 weeks later). In this circumstance, the best overall response can be interpreted as in Table 3.'

Table 3 of above-mentioned paper [1] is reported below and will be used to derive confirmed Best Overall Responses. In this study a minimum SD duration of 6 week will be used as criterium to confirm SD as Best Overall Response.

| Overall response<br>First time point | Overall response<br>Subsequent time point | BEST overall response |
|---|---|---|
| CR | CR | CR |
| CR | PR | SD, PD or PR <sup>a</sup> |
| CR | SD | SD provided minimum criteria for SD duration met, otherwise, PI |
| CR | PD | SD provided minimum criteria for SD duration met, otherwise, PI |
| CR | NE | SD provided minimum criteria for SD duration met, otherwise NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | SD provided minimum criteria for SD duration met, otherwise, PI |
| PR | NE | SD provided minimum criteria for SD duration met, otherwise NI |
| NE | NE | NE |

CR = complete response, PR = partial response, SD = stable disease, PD = progressive disease, and NE = inevaluable.

Patients with non-target disease only, may have a time point response of NON-CR/NON-PD, these responses will be included in the count of SD.

Determinations of Best Overall Responses derived as described will be reviewed by Symphogen and PAREXEL on a patient by patient basis across time.

#### Unconfirmed BOR by RECIST v1.1:

Per RECIST 1.1 [1]: in cases where confirmation of complete or partial response is not required the Best response is defined as the best response across all time points (for example, a patient who has SD at first assessment, PR at second assessment, and PD on last assessment has a best overall response of PR). When SD is believed to be best unconfirmed response, it must also meet the protocol specified minimum time from baseline.


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

a If a CR is truly met at first time point, then any disease seen at a subsequent time point, even disease meeting PR criteria relative to baseline, makes the disease PD at that point (since disease must have reappeared after CR). Best response would depend on whether minimum duration for SD was met. However, sometimes 'CR' may be claimed when subsequent scans suggest small lesions were likely still present and in fact the patient had PR, not CR at the first time point. Under these circumstances, the original CR should be changed to PR and the best response is PR.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

Patients with non-target disease only, may have a time point response of NON-CR/NON-

PD, these responses will be included in the count of SD.

Documented objective response (OR) confirmed and unconfirmed, based on determination

of confirmed and unconfirmed best overall response (BOR) per RECIST v1.1.

Confirmed OR is defined as the percentage of patients who had confirmed CR or PR.

Unconfirmed OR is defined as the percentage of patients who had unconfirmed CR or PR.

'The duration of overall response is measured from the time measurement criteria are

first met for CR/PR (whichever is first recorded) until the first date that recurrent or

progressive disease is objectively documented (taking as reference for progressive

disease the smallest measurements recorded on study). '[1].

Duration of Response (weeks) = (Date of PD – Date of first CR/PR [whichever is first

recorded] + 1) / 7

Time to Progression (TTP)

Time to documented PD (based on radiological assessments) will be derived and expressed

in the unit of weeks. TTP is defined as the time from first dose of study drug until objective

tumor progression; TTP does not include deaths [3]. Based on this definition, PDs will be

counted as outcome; patients with last tumor assessment showing CR or PR or SD will be

censored at the time of last available tumor assessment per RECIST v1.1; patients who

died for any cause (including deaths of disease but with no documented PD) will as well

be censored at the time of last available tumor assessment per RECIST v1.1.


TTP (weeks) = (Date of PD – Date of first IMP infusion + 1) / 7

In this study, there is no planned survival status after discontinuation of study treatment,

therefore, progression-free survival is not calculated.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

• Disease control rate (DCR), based on determination of confirmed BOR per RECIST v1.1.

The DCR is defined as the percentage of patients who had confirmed BOR of CR, PR or

SD of at least 16 weeks. Definition of duration of TTP corresponds to SD duration; thus,

these times will be used to determine if a patient was in SD for at least 16 weeks.

• Changes in sum of diameters of target lesions from baseline to end of trial participation

For patients with measurable disease (i.e., with target lesions), absolute and percent

changes in the sum of diameters of target lesions from baseline to end of trial participation

will be calculated, the best change will be identified as largest reduction or smallest

increase.

3.2.1.2 Tumor Markers

Tumor Markers that are part of the trial site standard practices, as indicated by tumor type, are

evaluated at timepoints coinciding with the CT/MRI imaging studies.

3.2.2 Pharmacodynamic, Biomarkers and Immunogenicity

These variables include:

• Archival Tumor Tissue for EGFR, HER2 and HER3 expression level, only applicable to

patients included in Part 1

• Biomarkers: Potential biomarkers of interest include genes, gene transcripts, and proteins

of the HER family receptors and molecules of the mitogen-activated protein kinase

(MAPK) and phosphoinositide 3-kinase (PI3K) pathways involved in HER signaling.

Peripheral blood samples are taken at Screening (after confirmation of eligibility); end of

Cycle 2 (prior to dosing Cycle 3) or upon PD, whichever occurs first; EOT.


• Skin biopsy: All patients enrolled will undergo skin biopsies for evaluation of target-

engagement (EGFR and HER3). Skin biopsy will be performed at Screening (after

confirmation of eligibility), and end of Cycle 2 (prior to dosing Cycle 3) or upon PD,

TP-GDO-WW-133-01

**Project Document Effective Date:** 05 April 2019

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

whichever comes first. Sampling procedure after amendment 6.0 (protocol version 7.0)

was changed to Screening (after confirmation of eligibility) and Cycle 1, day 8 and Cycle

1 day 15.

• Tumor biopsy: Optional for Part 1 and required for Part 2, will be performed after

confirmation of eligibility at Screening, and end of Cycle 2 (prior to dosing Cycle 3) or

upon PD, whichever occurs first. Analysis of tumor biopsies will include target-

engagement (EGFR, HER2 and HER3) and may furthermore include proteins and genes

that are unknown or have not been included in the scientific hypotheses at the present time

of trial, but that, during the collection of data from this trial, may evolve as new candidate

genes and markers related to Pan-HER safety, efficacy, or mechanism of action.

• Immunogenicity (ADA): Analysis of ADA and residual serum levels of Pan-HER will be

performed at a central laboratory. ADA will be assessed at C1/D1, C2/D1, Prior to every

second cycle thereafter, EOT, 1M FUP.

3.2.3 Pharmacokinetic Variables

Serum concentrations of each of the 6 monoclonal antibodies (mAbs) that comprise Pan-HER will

support the PK endpoints of the trial. The serum concentrations may also be used in an exploratory

population PK analysis which will be reported separately from the clinical trial report.


PK blood sampling schedules are summarized in below tables (Table 11 and Table 12 from

Clinical Study Protocol).


Symphogen A/S Sym013-01

Table 11 Schedule of Pharmacokinetic (PK) Assessments: Q1W Dosing

| | | Cycle 1 | | | | Cycle 2 Onward | | | | ЕОТ | 1M<br>FUP |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Sampling Time Window | Window | D1-<br>D3 | D8 | D15 | D22 | D1 | D8 | D15 | D22 | | |
| Prior to SOI | - 4 h | X | X <sup>1</sup> | X <sup>1</sup> | X1. | $X^1$ | X1 | X <sup>1</sup> | X <sup>1</sup> | | |
| EOI | + 10 min | X | $X^1$ | X <sup>1</sup> | X | X <sup>1</sup> | Xi | $X^1$ | X <sup>1</sup> | | |
| EOI+2h | ±30 min | X | | | X | | | | | | |
| EOI+4h | ±30 min | X | | | X | | | | | | |
| EOI + 8 h <sup>2</sup> | ±90 min | X | | | X | | | | | | |
| EOI + 24 h | ±6 h | X | | | Х | | | | | | |
| EOI + 48 h | -12 h to + 24 h | X | | | х | | | | | | |
| During Visit | NA | | | | | | | | | X | X |

Abbreviations (in alphabetical order): D. day; EOI, End of Infusion, EOT, End of Treatment Visit; NA, Not Applicable; h, hour, min, minutes; 1M FUP, 1-Month Follow-up Visit; SOI, Start of Infusion

- 1) If Pan-HER dosing is delayed, only one PK sample should be taken during the visit.
- 2) Effective with Amendment 6, sampling at this timepoint is optional.

Table 12 Schedule of Pharmacokinetic (PK) Assessments: Q2W Dosing

| | | Cycle 1 | | | | Cycle 2 | | Cycle 3<br>Onward | | ЕОТ | 1M<br>FUP |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Sampling Time | Window | D1-<br>D3 | D8 | D15 | D22 | D1-<br>D3 | D15 | D1 | D15 | | |
| Prior to SOI | - 4 h | Х | | X <sup>1</sup> | | X | X1 | $\mathbf{X}^{1}$ | X <sup>1</sup> | | 1 |
| EOI | + 10 min | Х | | X¹ | | Х | X1 | $X^1$ | X1 | | |
| EOI+2h | ±30 min | X | | | | X | | | | | |
| EOI+4h | ±30 min | X | | | | X | | | | | |
| EOI + 8 h <sup>2</sup> | ±90 min | X | | | | X | | | | | |
| EOI + 24 h | ±6 h | X | | | | X | | | | | |
| EOI + 48 h | -12 h to + 24 h | X | - | | | X | | | | | |
| During Visit | NA | | X | | X | | | | | X | X |

Abbreviations (in alphabetical order): D. day; EOI, End of Infusion, EOT, End of Treatment Visit; NA, Not Applicable; h, hour; min, minutes; 1M FUP, 1-Month Follow-up Visit; SOI, Start of Infusion

- 1) If Pan-HER dosing is delayed, only one PK sample should be taken during the visit.
- 2) Effective with Amendment 6, sampling at this timepoint is optional.

The PK endpoints with Q1W dosing will be derived based on the concentration time curves of Pan-HER after the first and fourth infusion of Pan-HER.

The PK endpoints with Q2W dosing will be derived based on the serum concentration time curves of Pan-HER after the first and third infusion of Pan-HER.

TP-GDO-WW-133-01 CONFIDENTIAL Project Document Version No. Final 1.0
Effective Date: 05 Sep 18
Related to: SOP-GDO-WW-019


Symphogen A/S Sym013-01

The planned PK endpoints are listed in Table 13 of Clinical Study Protocol.

The data may not allow for derivation of all endpoints for all mAbs, patients and occasions.  $C_{max}$ ,  $C_{EOI}$ ,  $C_{trough}$  and  $T_{max}$  will be derived from observed data while  $AUC_{\tau}$ ,  $AUC_{\tau 0}$ ,  $AUC_{norm, \tau}$ ,  $CL_{S}$ ,  $CL_{SS}$ ,  $V_{S}$ ,  $V_{SS}$ , and  $T_{\frac{1}{2}}$  will be estimated using non-compartmental methods and actual time points.

Table 13 Pharmacokinetic (PK) Endpoints, Definitions and Derivations

| Symbol | Definition and derivation |
|---|---|
| C <sub>trough</sub> | Trough concentration (i.e. concentration of Pan-HER measured pre-infusion) |
| $\mathrm{AUC}_{	au}$ | Area under the concentration-time curve in a dosing interval (i.e. from time zero (end of infusion) up to 168 hours). AUC $_{\tau}$ will be calculated using the linear trapezoidal method and interpolated in case of measurements after 168 hours, or extrapolated using terminal rate constant and the last quantifiable concentration |
| $\mathrm{AUC}_{	au0}$ | Area under the concentration-time curve from start of infusion up to 168 hours. $AUC_{\tau0}$ will be calculated similar to $AUC_{\tau}$ |
| AUC <sub>norm</sub> , τ | Dose normalized area under the concentration-time curve in a dosing interval, calculated as AUC $_{\tau}$ divided by the dose infused |
| C <sub>max</sub> | Maximum concentration |
| $T_{\text{max}}$ | Time to reach maximum concentration |
| C <sub>EOI</sub> | Concentration at End of Infusion |
| $\lambda_{\rm z}$ | Terminal rate constant (negative of the slope of an In-linear regression of the un-weighted data considering the terminal phase of the concentration-time curve $\geq$ limit of quantification). $\lambda_z$ is not an endpoint, but is used for derivation of endpoints |


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

Symphogen A/S Sym013-01

| Symbol | Definition and derivation |
|---|---|
| T1/2 | Terminal elimination half-life, calculated as $ln(2)/\lambda_z$ |
| $\mathrm{CL}_{\mathrm{S}}$ | Clearance after first dose, calculated as Dose/AUC <sub>inf</sub> for C1/D1, where AUC <sub>inf</sub> will be calculated as the sum of the area from time zero to time of last quantifiable concentration, $t_z$ , and the area from $t_z$ to infinity. The second area will be estimated using the observed concentration at $t_z$ and the terminal rate constant |
| CL <sub>SS</sub> | Clearance after $3^{rd}/4^{th}$ dose, calculated as Dose/AUC <sub><math>\tau</math></sub> |
| V <sub>S</sub> | Volume of distribution during the terminal phase after first dose $(CL_S/\lambda_z)$ |
| V <sub>SS</sub> | Volume of distribution during the terminal phase after $3^{rd}/4^{th}$ dose $(CL_{SS}/\lambda_z)$ |

#### 3.2.4 Safety Variables

The following safety endpoints will be assessed:

- Dose-Limiting Toxicities Evaluation
- (S)AE Survey
- Prior and concomitant medications (medications and/or treatments taken other than Pan-HER)
- Laboratory assessments (biochemistry, hematology, urinalysis, and coagulation)
- Pregnancy test
- 12-lead electrocardiogram (ECG)

Symphogen A/S Sym013-01

- Echocardiogram (ECHO) or Multi-Gated Acquisition (MUGA) Scan
- Vital Signs and Body Measurements
- Physical Examination
- Eastern Cooperative Oncology Group (ECOG) performance status (PS) score

#### 3.2.4.1 Dose Limiting Toxicity

A DLT is defined as any of the following toxicities that occur during the DLT-observation period, if considered related (causality rating of possibly, probably, or related) to Pan-HER:

- 1. Grade 3 non-hematologic toxicity regardless of duration, with the exception of:
  - a. Grade 3 nausea, vomiting, diarrhea, or fatigue lasting ≤2 days with best supportive care
  - b. Grade 3 asymptomatic electrolyte abnormality that is not considered clinically significant by the Investigator and that is controlled with medical therapy
- 2. Grade 4 non-hematologic toxicity, with the exception of:
  - a. Grade 4 asymptomatic electrolyte abnormalities that is not considered clinically significant by the Investigator and that is controlled with medical therapy
- 3. Neutropenia that is:
  - a. Grade 3-4 febrile neutropenia
  - b. Grade 4 and sustained (i.e., ANC  $< 0.5 \times 10^9 / L [500 / mm^3]$ , duration > 5 days)
- 4. Thrombocytopenia that is
  - a. Grade 3 with clinically significant hemorrhage
  - b. Grade 4 (platelets  $<25 \times 10^9/L$  [25,000/mm<sup>3</sup>])
- 5. AST/ALT elevation >3×ULN with bilirubin elevation >2×ULN without evidence of cholestasis that cannot be explained by factors not related to Pan-HER

TP-GDO-WW-133-01 CONFIDENTIAL Project Document Version No. Final 1.0 Effective Date: 05 Sep 18 Project Document Effective Date: 05 April 2019 

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

6. Evidence of cardiac toxicity as defined by either:

a. ≥16% absolute decrease in LVEF from baseline, or

b. LVEF below the institutional lower limit of normal and ≥10% absolute decrease in

LVEF from baseline

7. Inability to complete Cycle 1 at the assigned dose due to  $\geq$  Grade 3 toxicity

8. Treatment delays  $\geq$ 2 weeks from the scheduled next dose due to  $\geq$  Grade 3 toxicity

DLT events (Yes / No) are collected in CRF as well as date of assessment, DLT description and

AE Reference.

The decision to dose-escalate will be based on close monitoring of safety during the observation

period for DLTs, defined as the initial 28-day period (±2 days) from first treatment of Pan-HER

(i.e. Cycle 1) and including 7 days for Q1W or 14 days for Q2W of follow-up from the last dose

of Cycle 1.

A minimum of 4 infusions of Pan-HER (Q1W dosing) or 2 infusions of Pan-HER (Q2W dosing)

must have been administered at the assigned dose for a patient to have completed the DLT-

observation period.

3.2.4.2 Adverse Events

<u>Definitions</u>

An Adverse Event (AE) is any untoward medical occurrence in a patient or a clinical investigation

patient administered a pharmaceutical product, and which does not necessarily have a causal

relationship with this treatment. An AE can therefore be any unfavorable and unintended sign

(including an abnormal laboratory finding), symptom, or disease temporally associated with the

use of an IMP, whether or not considered related to the IMP.

Treatment-emergent AEs are events that occur on or after first dose of the study medication or a

worsening in severity of a preexisting condition occurring on or after first dose of the study


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

medication (a pre-existing is a condition that is present before the AE recording period starts and

is noted on the medical history/physical examination form).

An IRR is defined as an AE occurring during the Pan-HER infusion and up to 2 hours after the

end of infusion (EOI), which is assessed by the Investigator as possibly, probably, or related to

Pan-HER; IRRs (Yes/No) will be captured in CRF.

AE duration will be derived as AE duration = (AE end date - AE onset date +1); in case of AE

ongoing, the date of last contact with the patient will be used as AE for the scope of derive the AE

duration.

An SAE is an AE that meets one or more of the following outcome criteria:

• Results in death

• Is life-threatening (patient is at immediate risk of death at the time of the event; it does not

refer to an event which hypothetically might cause death if it was more severe)

• Requires in patient hospitalization (formal admission to a hospital for medical reasons) or

prolongation of existing hospitalization

• Results in persistent or significant disability/incapacity

• Results in a congenital anomaly/birth defect

• Is medically important (Medically important events may not be immediately life-

threatening or result in death or hospitalization but may jeopardize the patient or may

require intervention to prevent one of the other outcomes listed in the definition above)

All AEs will be recorded from signing of informed consent for participation in the trial. The

recording period ends at the time of the 1M FUP Visit.

All referenced toxicity grading within this protocol will be according to the CTCAE v4.03. If the

severity of an AE is not specifically graded by the CTCAE guidance document, the Investigator

should use the general definitions of Grades 1 to 5 as per the following, and use his/her best medical

judgment to describe the severity of the AE:

Symphogen A/S Sym013-01

• Grade 1: Mild

• Grade 2: Moderate

• Grade 3: Severe

• Grade 4: Life-threatening or disabling

• Grade 5: Death caused by the event

Changes in severity of AEs will be recorded.

AEs will be assessed for causal relationship to the IMP. The causal relationship of an AE to the IMP, Pan-HER, will be rated as follows:

• Not Related (The AE is not related to the IMP)

• Unlikely Related (The AE is considered not related to the IMP)

• Possibly Related (The AE might not be related, but possibility cannot be ruled out with certainty and therefore would be considered related)

 Probably Related (It has been determined with a high degree of certainty that the AE is associated with administration of IMP)

• Related (The AE is related to the IMP)

Outcome of the AE will be assessed utilizing one of the following terms:

Recovered

• Recovered with sequelae (if recovered with sequelae, specify sequelae)

Not recovered

Fatal

• Unknown

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

Handling of partial AE onset and end date

Any AEs with incomplete start and end dates will be treated as follows:

Adverse events with completely unknown onset date will be considered as treatment-emergent;

for the scope of AE duration derivation, these AE will be considered as occurred the day of

first IMP infusion.

Adverse events with unknown start day and month but with known start year will be

considered:

o as treatment-emergent if the start year coincides or is after the first dosing year; for

the scope of AE duration derivation, these AE will be considered as occurred the

day of first IMP infusion if the start year coincides with first dosing year, as

occurred on 1st January otherwise (i.e. in case the start year is after the first dosing

year)

o as non-treatment emergent if start year is before the first dosing year; for the scope

of AE duration derivation, these AE will be considered as occurred on 1<sup>st</sup> January.

Adverse events with unknown start day but with known start month and year will be

considered:

o as treatment-emergent if the start month and year coincide or are after the month

and year of first dosing; for the scope of AE duration derivation, these AE will be

considered as occurred the day of first IMP infusion if the start month and year

coincides with first dosing month and year, as occurred on 1st day of the month

otherwise (i.e. in case the month and year is after the month and year of first dosing)

o as non-treatment emergent if start month and year is before the month and year of

first dosing; for the scope of AE duration derivation, these AE will be considered

as occurred on 1st day of the month.

Adverse events with completely unknown end date will be considered as ended on the day of


last contact with the patient).

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

Adverse events with unknown end day and month but with known end year:

o if the AE end year if before the year of last contact with the patient, AE will be

considered as ended on 31th December.

o if the AE end year coincide with the year of last contact with the patient, AE

will be considered as ended on day of last contact with the patient.

o If AE end year is after the year of last contact with the patient, for the scope of

derive the AE duration the date of last contact with the patient will be used as

AE end date.

Adverse events with unknown end day but known end month and end year:

o if the AE end month and year are before the month and year of last contact with

the patient, AE will be considered as ended on last day of the month.

o if the AE end month and year are coinciding with the month and year of last

contact with the patient, AE will be considered as ended on last day of last

contact with the patient.

o If AE end month and year are after the month and year of last contact with the

patient, for the scope of derive the AE duration the date of last contact with the

patient as AE end date.

Adverse events with completely or partial unknown start and end dates will be shown as not known

(NK), for the respective unknown part, in the listings.

3.2.4.3 Clinical Laboratory and Pregnancy Test

Hematology panel (complete blood count with differential, ANC, and platelet count): at

Screening, Cycle 1 (weekly prior to dosing if on dosing day, Day 3. Note: Does not need

to be performed prior to C1/D1, if performed during screening  $\leq$ 7 days from C1/D1), each

cycle thereafter (Day 1 and 15 prior to dosing), EOT, 1M FUP, and as clinically indicated.


**Project Document Effective Date**: 05 April 2019


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

• Biochemistry panel (sodium, potassium, chloride, bicarbonate or carbon dioxide, blood

urea nitrogen (BUN), creatinine, glucose, bilirubin [total and direct], AST, ALT, ALP,

calcium, magnesium, phosphorus, albumin, total protein, uric acid, amylase, lipase, and

creatine kinase): at Screening, Cycle 1 (weekly prior to dosing if on dosing days, Day 3.

Note: Does not need to be performed prior to C1/D1, if performed during screening ≤7

days from C1/D1), each cycle thereafter (Day 1 and 15 prior to dosing), EOT, 1M FUP,

and as clinically indicated.

• Coagulation panel (PT, PTT and INR): at Screening, Cycle 1 (Day 1 and 15 prior to dosing.

Note: Does not need to be performed prior to C1/D1, if performed during screening ≤7

days from C1/D1), each cycle thereafter (Day 1 prior to dosing), EOT, 1M FUP, and as

clinically indicated.

• Urinalysis (specific gravity, pH, protein, glucose, ketones, occult blood, leukocyte

esterase, nitrite, bilirubin, and urobilinogen): at Screening, Cycle 1 (Day 1 and 15 prior

to dosing. Note: Does not need to be performed prior to C1/D1, if performed during

screening ≤7 days from C1/D1), each cycle thereafter (Day 1 prior to dosing), EOT,

1M FUP, and as clinically indicated.

• Pregnancy test (serum human Chorionic Gonadotropin (β-hCG) at screening, urine β-

hCG thereafter, in women of childbearing potential): at Screening, EOT and as

clinically indicated.

3.2.4.4 Electrocardiogram

A 12-lead ECG will be performed on Screening, EOT, and as clinically indicated.

Parameters measured will include heart rate, PR, R-R, QRS, QT, and QTc intervals (calculated

by the Fridericia [QTcF] or Bazzett's [QTcB] correction formula). Clinical assessment

(abnormality as clinically significant or not clinically significant) will be performed.

3.2.4.5 Echocardiogram (ECHO) or Multi-Gated Acquisition (MUGA) Scan

Transthoracic echocardiogram (ECHO) or Multi-Gated Acquisition (MUGA) scan will be

performed at Screening, EOT, and as clinically indicated.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

> Vital Signs and Body Measurements 3.2.4.6

Vital signs, including temperature, heart rate, blood pressure, and body weight will be

monitored at Screening, prior to each dosing, EOT, 1-month FUP and as clinically indicated.

3.2.4.7 Physical Examination

Full physical examination at Screening to include evaluation of: general appearance, skin, head,

ears, eyes, nose, throat, neck/thyroid, chest/breasts, lungs, cardiovascular system, abdomen,

musculoskeletal system, pulses, lymph nodes, neurologic status and mental status.

Thereafter, a targeted physical examination may be performed as indicated: at Screening, Day

1 of each cycle prior to dosing, EOT, 1M FUP and as clinically indicated.

3.2.4.8 Eastern Cooperative Oncology Group (ECOG) performance Status (PS) score

ECOG PS will be assessed at Screening, Day 1 of each cycle (prior to dosing), EOT, 1M FUP and

as clinically indicated.

ECOG PS Score:

0=Fully active, able to carry on all pre-disease activities without restrictions

1=Restricted in physically strenuous activity but ambulatory and able to carry out work of

a light or sedentary nature e.g., light housework, office work

2=Ambulatory and capable of self-care, but unable to carry out any work activities. Up

and about more than 50% of waking hours

3=Capable of only limited self-care, confined to bed or chair more than 50% of waking

hours

4=Completely disabled. Cannot carry on self-care. Totally confined to bed or chair

5=Dead

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

STATISTICAL METHODS

**Data Quality Assurance** 

All tables, figures and data listings to be included in the report will be independently checked for

consistency, integrity and in accordance with standard PAREXEL procedures.

4.2 **General Presentation Considerations** 

**Baseline** 

'Baseline' is defined as the last available pre-treatment assessment, considering both scheduled

and unscheduled assessments.

Safety assessments at Cycle 1 Day 1 with no time of assessment (i.e. Vital Signs and Body

Measurements, ECOG PS, Physical Examination) are assumed to be taken pre-treatment.

**End of Treatment (EOT)** 

'End of Treatment' is defined as the first assessment on or after the last dose of study treatment,

considering both scheduled and unscheduled assessments.

**Unscheduled assessments** 

Unscheduled assessments will be presented in listings in chronological order.

Post Baseline unscheduled assessments (for Clinical Laboratory, ECG QTc, etc.) will be used for

determination of worst result (i.e. Maximum and Minimum post Baseline result) as well as the

maximal laboratory CTCAE grade if applicable; also, all post baseline tumor evaluation

assessments will be used to derive BOR.

Except considered as Baseline, EOT or worst result, unscheduled assessments will not be included


in summaries.


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

**Treatment Day** 

'Treatment Day' will be calculated relative to the date of C1/D1 as follow:

• assessments taken before the first infusion of IMP

Treatment Day = Assessment Date - First IMP infusion Date

• assessments after the first infusion of IMP

Treatment Day = Assessment Date - First IMP infusion Date + 1.

**Missing Data** 

In case of partially missing date of birth or date of diagnosis, the following rule will be applied: if

year and months are known but day is missing, then the day will be imputed as 15<sup>th</sup>; in case of only

year known, the day and month will be imputed as 15<sup>th</sup> June.

Specific rules for handling for missing efficacy assessments are detailed in section 4.10.1.3.

Methods for handling missing concomitant medication and adverse events dates are detailed in

sections 4.8 and 3.2.4.2 respectively.

Imputations will be used to derive parameters, in listings original data will be presented as

collected.

**Data Listing** 

All original and derived parameters for all consented patients will be listed.

All listings will include scheduled and unscheduled measurements.

Unless specified otherwise, data in listings will be presented by dose regimen (Q1W or Q2W),

dose group, patient, and visit (ordered by date and time within patient).

All listings will display the same number of decimals as in the source data. All raw data will be

reported exactly as provided.

Quantitative derived variables (e.g. Duration of Response, Time to Progression, Actual Treatment

duration) will be shown with 1 decimal place (d.p.) precision.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

The data for the patients who consented but for any reason did not receive any dose of study drug

(including screening failures) will be also listed but with a label of "and a footnote to flag these.

Efficacy, Exposure and PK/PD Data Listing will be based on Full Analysis Set.

**Tables and Descriptive Statistics** 

Unless specified otherwise all tables and statistics will be presented using the FAS.

Evaluation of DLT will not be based on FAS but on DLT Analysis Set.

Unless specified otherwise summary tables and figures will be presented by dose regimen (Q1W

or Q2W), dose group, and visit (where applicable); also, overall summaries will be shown for the

two-dosage regimen and for all patients pooled together. In general, summary tables will be

structured in three parts: first part will summarize overall results obtained in the two dose regimens

Q1W, Q2W and in all patients pooled together; second part will display all dose groups within the

dosage regimen Q1W; third part will display all dose groups within the dosage regimen Q2W.

In general, for variables showing multiple possible categories, these will be displayed with

following the within variable logic criteria, for example: ECOG categories will be displayed from

0 and going to grow; where such a logic criterium does not exist (example: gender, ethnicity, SOC,

PT), categories will be displayed by descending frequencies based on the overall all patients pooled

together. In the end, the order used to show categories within variables should be the same in the

three parts of each table.

Unless otherwise stated, continuous data will be summarized using descriptive statistics including:

number of non-missing observations (n), arithmetic mean, standard deviation (SD), median,

minimum, and maximum.

Categorical data will be summarized in terms of the number of patients providing data at the

relevant time point (n), frequency counts and percentages. Any planned collapsing of categories

will be detailed in the SAP text and the data displays. Percentages will be calculated using n as the

denominator. Changes from baseline in categorical data will be summarized using shift tables

where appropriate.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

The following rules will apply to all descriptive statistic displays, except the PK concentrations

and parameters that are reported in significant digits described in section 4.10.4.4 below, where d

denotes the decimal places in the original reported value:

n: 0 decimal places (d.p.)

Mean: d + 1 d.p.

Confidence Interval: d + 1 d.p.

SD: d + 2 d.p.

Median: d + 1 d.p..

Minimum: d.

Maximum: d.

Statistics in percentage: 1 d.p.

p-value: 4 d.p.

Except for p-value, a maximum of 3 decimal places will be displayed.

P-values greater than or equal to 0.001, in general, will be presented to three decimal places. P-

values less than 0.001 will be presented as "<0.001".

Details for reporting of statistical summaries specific to PK are detailed in section 4.10.1.4.

**Figures** 

If not otherwise specified, each figure will be presented separately for the two dose regimens (Q1W

and Q2W) with differentiate legend to discriminate the dose groups within the regimen; moreover,

an overall figure will also be presented with differentiate legend to discriminate the two dose

regimens. In the end, there will be three panel for each figure: first panel will show all patients,

second panel patients in Q1W regimen, third panel patients in Q2W regimen.


All figures will be produced in black and white.

**Project Document Effective Date**: 05 April 2019


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

Specification for PK figures will be detailed in section 4.10.4.1.

4.3 Software

The tables, listings, figures and any non-descriptive statistical analysis will be produced using

SAS® Software (Version 9.3 or higher). The REPORT procedure (SAS PROC Report) will be

used to produce all tables and listings; SAS/GRAPH will be used to produce all figures.

All tables, listings, and graphs will be produced to landscape orientation using Courier New 9pt

font and will be incorporated into a MS Word document as a (RTF) rich text file (margins on

standard A4: Margins (top, left, right, and bottom) 2.54 cm.

4.4 Study Patients

**4.4.1** Disposition of Patients

The patient disposition including the date the informed consent was signed, date of last infusion

of study drug and the primary reason for discontinuation of study treatment will be listed.

Moreover, the number of patients who consented to the study, were exposed to study treatment

and primary reason for end of treatment will be summarized.

Those patients who did not meet the eligibility criteria or were screen failures will be listed.

A listing of patients included into each of the analysis set will be presented, related summary

statistics will be provided.

A clear accounting of the disposition of all patients who enter the study will be provided, from

screening to study completion.

4.4.2 Protocol Deviations

A protocol deviation is any change, divergence, or departure from the study design or procedures

of a study protocol. All protocol deviations will be listed by patient. All protocol deviations will

be discussed during Data Review Meeting (DRM) and addressed with the "final" classification

together their overall effect on a patient, as well, assignment of each patient to the analysis sets

will be decided. During DRM, all protocol deviations and their possible impacts will be discussed

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

between PAREXEL and Symphogen and will be assessed as "minor" or "major". Major protocol

deviations and protocol deviations affecting primary analyses can lead to the exclusion of a patient

from the analysis sets. Reasons for excluding patients from any analysis set will be reported and

described in the DRM Report that will be finalized before database hard lock and signed off by all

relevant scientific experts.

4.5 Analysis Sets

Two analysis sets will be defined in accordance with the consolidated ICH E9 GCP guidelines.

The Full Analysis Set (FAS) will comprise all enrolled patients who have received at least one

dose of Pan-HER. The FAS will be used for evaluation of all endpoints except evaluation of DLTs.

The patients in the FAS will contribute to the analyses as allocated to treatment (patients will be

reported below the regimen and dosage actually received). For the evaluation of PK endpoints,

patients, full profiles, or single measurements can be excluded from the analyses with justification.

The decision of excluding patients, full profiles, or part of profiles will be described in the clinical

trial report (CTR).

The DLT Analysis Set will comprise all patients in the FAS enrolled in Part 1, except patients who

did not complete Cycle 1 for reasons other than drug toxicity. The DLT Analysis Set will be used

for evaluation of DLTs and the MTD or lack thereof.

4.6 Demographics and Baseline Characteristics, Disease History and Prior Cancer


**Therapies** 

The following demographic and baseline variables will be recorded:

• Date of informed consent

Date of Birth

• Gender, Race and Ethnicity

Height

Weight at screening and baseline

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

Stage at initial diagnosis and current stage

• Screening and baseline ECOG PS (categories)

• Disease history and diagnosis (Site of primary tumor, Date of initial diagnosis, Sites of

metastases, Date of most recent progression)

• Prior cancer therapies including prior surgical treatment [yes/no], prior radiation therapy

[yes/no] and prior systemic therapies, Prior anti-EGFR treatments [yes/no] and Responder

to prior anti-EGFR treatments [Positive/Negative], Prior HER2 therapies [yes/no] and

Responder to prior HER2 therapies [Positive/Negative]

Age at consent in years will be derived as (Year of informed consent signed – Year of date of birth)

+ 0 if the month and day of informed consent signed >= the month and day of date of birth, else +

1. The following age classes will be as well derived: < 65 years; 65 - <75 years; 75 - <85 years;

85 years or older.

BMI at baseline will be calculated as Weight [kg] / (Height [m])<sup>2</sup>

Time since initial diagnosis will be derived as (Year of informed consent signed – Year of initial

diagnosis) + 0 if the month and day of informed consent signed >= the month and day of initial

diagnosis, else + 1.

Number of sites with metastases will be derived by counting all sites with metastases.

Prior systemic therapies for cancer will be counted by regimen and summarized as 0, 1, 2, 3, 4+

for each patient.

Regimens containing anti-EGFR or HER2 drugs will be identified.

Demographic and baseline characteristics, Disease History and Prior Cancer Therapies will be

listed.

Listing of Systemic Therapies will be reviewed by Symphogen and PAREXEL and regimens with

anti-EGFR or HER 2 treatments will be flagged, data should then match with answers collected in

CRF for prior anti-EGFR treatments [yes/no] and Prior HER2 therapies [yes/no]; cases of


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

mismatch will be queried; any unsolved case of mismatch will be reviewed by on a patient by

patient basis.

Descriptive continuous statistics will be presented for:

Demographic and baseline characteristics (including age, height, weight and BMI)

Disease History information (including Time since initial diagnosis [years]).

The frequency and percentage of patients will be tabulated for:

Demographic and baseline characteristics categorical variables (including gender, race, and

ethnicity);

Disease History information (including ECOG PS, Site of primary tumor, number and sites

of metastases, EGFR and HER2 results [positive/negative])

Prior Cancer Therapies for current malignancy (including prior surgical treatment [yes/no],

prior radiation therapy [yes/no], number of prior systemic therapies [0, 1, 2, 3, More than

3], Prior anti-EGFR treatments [yes/no] and Responder to prior anti-EGFR treatments

[yes/no], Prior HER2 therapies [yes/no] and Responder to prior HER2 therapies [yes/no]).

The stage at initial diagnosis and current stage will only be listed.

4.7 **Medical History and Concomitant Illnesses** 

Medical history is assessed at screening and include prior and ongoing medical illnesses and

conditions and prior surgical procedures not related to the primary diagnosis.

Medical History terms will be coded using MedDRA, 19.1. Medical History terms will be listed.

4.8 **Prior and Concomitant Medications** 

Medications are all prescription medications, over-the-counter medications, or alternative

therapies registered from screening through 30 days after the last dose of study drug. Medications

will be listed (excluding those taken prophylactically for Pan-HER reactions).


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

Medications will be coded using the World Health Organization Drug Dictionary drug (WHODD,

September 2016 and will be presented by WHODD Anatomical-Therapeutic-Chemical (ATC)

therapeutic classification and preferred term (PT).

Medications and treatments administered prior to the first infusion of study drug which stopped

prior to first infusion of study drug will be considered as prior medications and flagged in the

listing.

Medications and treatments which started before, on or after the first infusion of study drug and

which stopped after first infusion of study drug (including medications and treatments which

stopped the day of first infusion) will be considered as concomitant medications.

If medication start and/or stop dates are missing or partial, the dates will be compared as far as

possible with the date of first dose of study medication. Medications will be assumed to be

concomitant, unless there is clear evidence (through comparison of partial dates) to suggest that

the medication stopped prior to the first dose of study medication. If there is clear evidence to

suggest that the medication stopped prior to the first dose of study medication, the medication will

be assumed to be Prior.

Prophylactic treatment for Pan-HER related reactions and pre-medication for Pan-HER infusions

will be listed separately.

Concomitant procedures performed during the study will be collected and listed.

4.9 Treatment Exposure and Compliance

Data of study drug infusion including dose reduction and interruption information, patient drug

administration irregularities (dose reduction and interruption) and infusion related reaction will be

listed.

Duration of the Pan-HER exposure, treatment duration, actual number of doses, planned total dose,

actual total dose and Relative Dose Intensity (RDI) will be derived as follow:


• Duration of exposure (days) = (last dose date - first dose date +1)

• Actual Treatment duration (weeks) =

Symphogen A/S Sym013-01

(last dose date - first dose date + 7) / 7 for weekly dose (i.e. dose regimen Q1W), or (last dose date - first dose date + 14) / 7 for biweekly dose (i.e. dose regimen Q2W)

- Number of treatment cycles initiated (i.e. at least one infusion for the cycle)
- Number of treatment cycles completed (i.e. all cycle infusions were received by the patient)
- Planned total number of doses for Q1W = (Date of last dose Date of first dose +1) / 7 rounded up to integer
- Planned total number of doses for Q2W = (Date of last dose Date of first dose +1) / 14
   rounded up to integer
- Planned total dose = Planned dose \* Planned total number of doses
- Planned treatment duration (weeks) for Q1W = Planned total number of doses  $\times$  1
- Planned treatment duration (weeks) for Q2W = Planned total number of doses  $\times$  2
- Relative dose intensity (RDI)

RDI (%) = 
$$100 \times \frac{\text{Sum of all received dose / Duration of exposure (days)}}{\text{Total planned dose / (Planned treatment duration (weeks)x7)}}$$

whereas the total planned dose (mg/kg) and planned dose duration are calculated based on the number of doses of the study medication a patient had received at the initially planned dose (mg/kg) for the cycle according to the planned dosing schedule.

Example, if a patient received 8 bi-weekly (i.e. dose regimen Q2W) doses of a study medication with a loading dose of 12 mg/kg and rest 9 mg/kg, with 1 dose reduction from 9 mg/kg to 6 mg/kg starting at week 14 and 1 week delay and at week 16, then

RDI (%) = 
$$100 \times \frac{(12 + 5 \times 9 + 2 \times 6) / 119}{(12 + 7 \times 9) / 112} = 86.6\%$$

The number of initiated and completed cycles of taking Pan-HER will be summarized both as categoric (0, 1, 2, 3, 4, 5, >5) and continuous parameter.


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 Project Document Version No. Final 1.0 Project Document Effective Date: 05 April 2019 

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

Duration of the Pan-HER exposure will be summarized as actual treatment duration (weeks) and

actual number of doses. RDI will be summarized both as categoric (> 100%; 90 % - 100 %; 80 %

- < 90%; 70 % - < 80%) and continuous parameter. Swimmer Plot will be presented showing

Treatment Duration together with Tumor Response data.

Number of patients who had dose reduction (Any, 1, 2, 3+ times) and dose interruption (Any, 1,

2, 3+ times)) will be summarized.

4.10 Efficacy Evaluation

4.10.1 Analysis and Data Conventions

No formal testing of hypotheses has been planned in this study. Therefore, no formal sample size

calculations were performed.

Two-sided Confidence Intervals will be presented with  $\alpha$ =0.05 (95% CI).

4.10.1.1 Multi-center Studies

There will not be any adjustment for study centers, subgroup analysis based on study centers are

not planned.

4.10.1.2 Adjustments for Covariates

No statistical models will be provided for the analysis of Study Endpoints. All study analyses will

be descriptive and will be seen from an exploratory perspective. No adjustment for covariates is

then expected.

4.10.1.3 Handling of Dropouts or Missing Data

Efficacy data that are reported as missing will be excluded from all descriptive and non-descriptive

data analysis. There will be no imputation of missing efficacy data.

For general rules about handling of missing data refer to section 4.2.

4.10.1.4 Multiple Comparisons/Multiplicity

Not Applicable.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

4.10.1.5 Interim Analyses

No formal interim analysis is planned.

All relevant safety, PK and toxicity data will be reviewed on an ongoing basis throughout the trial,

especially at various decision points for dose escalations and expansion.

4.10.1.6 Examination of Subgroups

Tumor Type will be used as a subgroup to summarize some study endpoints or as stratification

factor in certain graphics as appropriately described in the text of this SAP. Tumor type

categorization will be based on primary tumor site which may also be combined with tumor

histology.

4.10.2 Analysis of Efficacy Variable(s)

All statistical analysis of the efficacy endpoints will be presented using the FAS.

4.10.2.1 Anti-Tumor Response according to RECIST v1.1

The following anti-tumor response endpoints will be measured in Part 1:

• Confirmed and unconfirmed BOR by RECIST v1.1 will be listed and summarized by dose

regimen and dose level received using frequency distribution for the categories CR, PR,

SD, PD, and Not Evaluable.

Number and percentage of patients with documented confirmed and unconfirmed OR will

be summarized by dose regimen and dose level using frequency distribution with the

corresponding 95% exact Clopper-Pearson Confidence Intervals (CI) for binomial

proportion. All documented ORs will be listed including duration (weeks) of response.

• Patients in DCR will be listed and summarized by dose regimen and dose level using


frequency distribution with the corresponding 95% exact Clopper-Pearson Confidence

Intervals (CI) for binomial proportion.

• Time to Progression (TTP)

**Project Document Effective Date:** 05 April 2019


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

The median TTP, as well as 26 weeks and 52 weeks TTP rates and the corresponding 95%

CIs will be estimated using the product-limit method and presented using a Kaplan-Meier

plot. Number and percent of censored patients will be presented, also number and percent

of patients censored for death will be presented.

Changes in sum of diameters of target lesions from baseline to end of trial participation

Changes in the sum of diameters of target lesions from baseline to end of trial participation

will be listed as percentage and absolute value, the best change (i.e., largest reduction or

smallest increase) will be identified and presented using summary table and plotted with a

waterfall plot. Change in sum of diameters will also be presented by primary tumor type.

Results of the tumor evaluation by CT/MRI for target lesions, non-target lesions and

timepoint tumor response will be listed, as well as derived target and non-target time point

responses.

4.10.2.2 Tumor Markers

The date of the tumor evaluation and all test results will be listed.

4.10.3 Pharmacodynamic, Biomarkers and Immunogenicity

4.10.3.1 Pharmacodynamic, Biomarkers, Immunogenicity (ADA) and Archival Tumor

Exploratory analysis may be conducted according to the study exploratory objectives based on the

available pharmacodynamic data.

Potential biomarkers of interest include genes, gene transcripts, and proteins of the HER family

receptors and molecules of the mitogen-activated protein kinase (MAPK) and phosphoinositide 3-

kinase (PI3K) pathways involved in HER signaling.

Results of pharmacodynamic biomarkers taken from blood samples will be listed. Blood sample

results for anti-drug antibody will be listed. Cancer Gene Mutations will be listed as well.


Exploratory analysis of the biomarker profiles might be performed.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

4.10.3.2 Skin Biopsy

The location of the skin biopsy, the date taken, and expression results of EGFR and HER3 and

proliferation marker Ki67 will be listed.

EGFR and HER3 receptor down modulation and changes in Ki67 in skin biopsies, measured by

percentage and nominal change in target expression from baseline to end of Cycle 2 or PD

(whichever comes first) in skin samples will be presented by tumor type using descriptive statistics.

After protocol amendment 6, (version 7.0), EGFR and HER3 receptor down modulation in skin

biopsies, measured by percentage and nominal change in target expression from baseline to Cycle

1 day 8 and Cycle 1 day 15 in skin samples will be presented by trial part and tumor type using

descriptive statistics, scatter plots of values at Cycle 1 day 8 and Cycle 1 day 15 versus baseline

may also be produced.

4.10.3.3 Tumor Biopsy

The date of the tumor biopsy, the tumor site, expression results of EGFR, HER2, and HER3 and

Ki67 satining will be listed. EGFR, HER2 and HER3 receptor down modulation and changes in

Ki67 in tumor biopsies (may not be available in Part 1), measured by percentage and nominal

difference in target expression from baseline to end of Cycle 2 or PD (whichever comes first) in

tumor biopsy samples will be presented by tumor type using descriptive statistics including scatter

plots of values at end of Cycle 2 versus baseline.

4.10.4 Pharmacokinetics

4.10.4.1 Pharmacokinetic Concentrations

Serum concentrations for each of the six monoclonal antibodies in Pan-HER will be listed by mAb,

dose schedule, dose group, patient, actual time relative to dosing, scheduled time and time

deviation from scheduled time. The unit for the concentrations will be µg/mL.


Patient profiles serum concentrations vs. time points for each mAb will be plotted by dose schedule

and dose group.

The following definitions are used for PK plots and tables:

**Project Document Effective Date:** 05 April 2019

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

• First profile for weekly: all PK points from Cycle 1 Day 1 to Cycle 1 Day 8 (pre-dose)

• 2<sup>nd</sup> profile for weekly (4<sup>th</sup> dose): all PK points from Cycle 1 Day 22 to Cycle 2 Day 1 (pre-

dose)

• First profile for biweekly: all PK points from Cycle 1 Day 1 to Cycle 1 Day 15 (pre-dose)

2<sup>nd</sup> profile for biweekly (3<sup>rd</sup> dose): all PK points from Cycle 2 Days 1to Cycle 2 Day-15

(pre-dose).

• Dosing/sampling occasions for weekly dosing: Week 1, 2, 3, 4, 5, 6 etc., EOT, 1MFUP

• Dosing/sampling occasions for biweekly dosing: Week 1, 3, 5, 7, 9 etc., EOT, 1MFUP

Peaks: serum concentration for each mAb assessed at EOI for each dosing occasion

• Troughs: serum concentrations for each mAb assessed prior to SOI for each dosing

occasion

Violations of scheduled sampling will be reviewed on a patient by patient basis by Symphogen

and PAREXEL. Following data review by Symphogen's pharmacokinetic expert, data points may

be excluded from mean calculations and parameter calculation based on the below criteria:

• Individual outlying data points which are markedly deviating from the preceding and

following time points

Data points or PK profiles which are not compatible with known physiological processess

underlying the PK properties

Unexpected events or protocol deviations documented in e.g. laboratory notes or in


protocol deviation reviews

Exclusions will be documented in the study files and the PC/PP files.

Following plots will be produced:


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

One panel per mAb, Dose Schedule and Dose group combination showing a profile for

each patient: Patient Profiles for concentration vs. Actual Time by Dose Schedule and

Dose Group (peak and trough for each dosing occasion) – Linear

One panel per mAb, Dose Schedule and Dose group combination showing a profile for

each patient: Patient Profiles for concentration vs. Actual Time by Dose Schedule and

Dose Group (peak and trough for each dosing occasion) Semi-log

One panel per patient with overlaid profiles of all six mAbs: concentration of the six mAbs

vs. Actual Time (peak and trough for each dosing occasion) – Semi-log

One panel per mAb, Dose Schedule and Dose group combination showing a profile for

each patient: Patient Profiles for concentration vs. actual time by Dose Schedule and Dose

Group (First and 2<sup>nd</sup> profiles) – Linear

One panel per mAb, Dose Schedule and Dose group combination showing a profile for

each patient: Patient Profiles for concentration vs. actual time by Dose Schedule and Dose

Group (First and 2<sup>nd</sup> profiles) – Semi-log

One panel per patient with overlaid profiles of all six mAbs vs. actual time (First and 2<sup>nd</sup>

profiles) – Semi-log

Above plots produced per mAb, Dose Schedule and Dose group combination will be composed

by one panel for each mAb; moreover, each panel will be composed by the following 7 sub-panels


Sub-panel a) all patients in q1w - 1mg/kg

Sub-panel b) all patients in q1w - 2mg/kg

Sub-panel c) all patients in q1w - 4mg/kg

Sub-panel d) all patients in q1w - 6mg/kg + P

Sub-panel e) all patients in q2w - 6mg/kg

Sub-panel f) all patients in q2w - 9mg/kg and 9mg/kg + P

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

Sub-panel g) all patients in q2w - 12mg/kg + P

Descriptive summary (n, arithmetic mean, SD, median, minimum, maximum, geometric means,

and CV% values) of serum concentrations of each of the six mAbs will be tabulated by dose

schedule, dose group and nominal sampling time. Following tables will be produced:

Summary of concentration for each of the six mAbs by Dose Group and Time Point (First and 2<sup>nd</sup>

profiles)

Summary of concentration for each of the six mAbs by Dose Group and Time Point (Peak and

trough for each dosing occasion)

The arithmetic and geometric means of the serum concentrations of each of the six mAbs vs.

nominal time points will be plotted by dose group with +/-1 standard deviation (for arithmetic

means). In figures of geometric means, error bars will be calculated using the following formula:

Exp (mean Ln +/- sd Ln) where 'sd Ln' denotes the standard deviation of the concentration values

on the log base 10 scale and 'mean Ln' denotes the arithmetic mean of the concentration values on

the log base 10 scale.

The following mean concentration vs. time plots will be produced:

Arithmetic Mean Concentration for each of the six mAbs vs. Planned Time Point by Dose

Group and Dose Schedule (First and 2<sup>nd</sup> profiles) – Linear

Geometric Mean Concentration for each of the six mAbs vs. Planned Time Point by Dose

Group and Dose Schedule (First and 2<sup>nd</sup> profiles) – Semi-log

Arithmetic Mean Peak and Trough Concentrations for each of the six mAbs vs. Planned Time

Point by Dose Group and Dose Schedule (peaks and troughs at all dosing occasions) -

Linear

Geometric Mean Peak and Trough Concentrations for each of the six mAbs vs. Planned Time


Point by Dose Group and Dose Schedule (peaks and troughs at all dosing occasions) –

Semi-log

**Project Document Effective Date**: 05 April 2019


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

4.10.4.2 Handling of Values Below the Limit of Quantification (BLQ)

Handling of values below the limit of quantification (BLQ) and missing data in listings and for the

calculation of descriptive statistics at each time point:

• At a time point where less than or equal to 50% of the values are BLQ, all BLQ values will

be set to the ½\*lower limit of quantification (LLOQ), and all descriptive statistics will be

calculated.

• At a time point where more than 50% of the values are BLQ, the mean, SD, geometric

mean and CV% will be set to Not Determined (ND). The max value will be reported from

the individual data, and the min and median will be set to BLQ.

• If all values are BLQ at a time point, no descriptive statistics will be calculated for that

time point. Not Applicable (NA) will be written in the field for SD and CV% and BLQ will

be written in fields for mean, geometric mean, min, median, and max.

• The number of BLQ values (n below LLOQ) will be reported for each time point.

4.10.4.3 Pharmacokinetic Parameters

Pharmacokinetic parameters for the first and second PK profile (as defined in 4.10.4.1) for each

patient and each monoclonal antibody will be derived by model-independent, non-compartmental

analysis (NCA) according to Symphogen's local procedures.

All derived serum PK parameters will be listed by mAb, dose schedule, dose group, patient, and

actual time point (Listing 16.2.6.2.1-2) and summarized descriptively by mAb, dose schedule and

group and day (Table 14.2.2.1-2). The following descriptive statistics will be presented for PK

parameters: n, arithmetic mean, SD, geometric mean, geometric CV% (calculated as:

gCV%=SQRT(exp(s<sup>2</sup>)-1)\*100; where s is the standard deviation of the log-transformed values),

median, minimum and maximum values.

4.10.4.4 Pharmacokinetic Analysis

Descriptive statistics of serum concentrations will be reported with the same precision as the source


data and serum concentrations.

Symphogen A/S Sym013-01

In addition to general continuous summary statistics presented in section 4.2, for PK parameters, geometric means with coefficient of variation (CV %) will be also summarized.

For drug concentrations and concentration-dependent pharmacokinetic parameters, the rules of data presentation are described in table below.

# Presentation of PK Parameters and Summary Statistics

| Typical | | | Minimum | Mean | | Geometric | CV |
|---|---|---|---|---|---|---|---|
| Variable | N | Digit rule | /Maximum | Median | SD | Mean | (%) |
| concentration | X | Significant digits | 3 | 4 | 4 | 3 | 3 |
| $C_{\text{max}}$ | X | Significant digits | 3 | 4 | 4 | 4 | 4 |
| $t_{\max}^*$ | X | Fixed decimal places | as raw data | as raw data | - | - | - |
| $\lambda_{\mathrm{z}}$ | X | Significant digits | 4 | 3 | 5 | 5 | 5 |
| $t_{1/2}$ | X | Significant digits | 3 | 3 | 4 | 4 | 4 |
| AUC <sub>(0-xx)</sub> | X | Significant digits | 3 | 3 | 4 | 4 | 4 |
| $AUC_{(0-\tau)}$ | X | Significant digits | 3 | 3 | 4 | 4 | 4 |

<sup>\*</sup> Mean and SD, geometric mean and CV will not be calculated for t<sub>max</sub>.

# 4.11 Safety Evaluation

All safety summaries will be based upon the FAS as defined in Section 4.5.

# 4.11.1 The DLT Analysis Set will be used for evaluation of DLTs Dose Limiting Toxicities (DLT)

All DLT events will be listed. Presence and absence of DLTs will be presented by regimen and dose in the order of date of first dose.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

4.11.2 Adverse Events

The AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 19.

1.

TEAEs will be presented by MedDRA System Organ Class (SOC) and Preferred Term (PT). In all

AE summary tables, SOCs and PTs will be presented in the order of descending frequencies as

detailed in section 4.2. AE frequency accounts for number and percent of patients who have a

specific SOC and PT as well as the worst grade, if there were multiple occurrences at different

toxicity grade, which was determined using CTCAE v4.03.

For purposes of the summary tables, AEs will be classified as either being related to study drug or

not related. AEs related to study drug will include AEs classified as 'Related', 'Probably Related'

or 'Possibly Related'. AEs not related to study drug will include AEs that are 'Unlikely Related'

or 'Not Related'.

All AEs will be listed. The AEs will be presented using summary tables including:

• Patient Overall Summary of TEAEs. This table will include following summaries:

o Any TEAEs

Any related TEAEs

Any Serious TEAEs

Any related Serious TEAEs

o Grade 3 or higher TEAEs

o Any Related Grade 3 or higher TEAEs

o Any TEAEs leading to Permanent Discontinuation of IMP

o Any Related TEAEs leading to Permanent Discontinuation of IMP

o Any TEAEs leading to interruption or Stop of study drug

Any Related TEAEs leading to interruption or Stop of study drug

Symphogen A/S Sym013-01

- O Any TEAEs with an outcome of reduction or delay of study drug
- o Any Relate TEAEs with an outcome of reduction or delay of study drug
- Any FATAL TEAEs
  - Fatal TEAEs within 30 days from last IMP infusion
  - Fatal TEAEs beyond 30 days from last IMP infusion
- TEAEs by Dose Group, SOC and PT
- Related TEAEs by Dose Group, SOC and PT
- TEAEs by Dose Group, SOC and PT and Worst CTCAE Grade
- Related TEAEs by Dose Group, SOC and PT and Worst CTCAE Grade
- Serious TEAEs by Dose Group, SOC and PT
- Related Serious TEAEs by Dose Group, SOC and PT
- TEAEs Leading to Withdrawal from Treatment by Dose Group, SOC and PT
- Related TEAEs Leading to Withdrawal from Treatment by Dose Group, SOC and PT
- Serious Adverse Events Key Patient Information (non TEAEs will be flagged)
- Adverse Events with Outcome of Death Key Patient Information (non TEAEs will be flagged)
- Adverse Events Leading to Discontinuation of Investigational Product Key Patient Information
- Adverse Events Leading to Dose Reduction Key Patient Information
- Adverse Events Leading to Dose Interruption- Key Patient Information
- Adverse Events Leading to Dose Stopped Key Patient Information

TP-GDO-WW-133-01 CONFIDENTIAL
Effective Date: 05 Sep 18
Related to: SOP-GDO-WW-019

Project Document Version No. Final 1.0 Project Document Effective Date: 05 April 2019


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

• Listing of Death (Deaths occurring within 30 days from last infusion of IMP will be

flagged.) (non TEAEs will be flagged)

4.11.3 Deaths, Serious Adverse Events, and Other Significant Adverse Events

Reporting of Deaths, Serious Adverse Events and other significant Adverse Events is described in

the above section 4.11.2.

4.11.4 Clinical Laboratory Evaluation

All clinical laboratory test results will be presented and summarized using the International System

of Units (SI units; Système International d'Unités). The original lab test units will be converted to

SI according to Young, D.S and Huth, E.J; 1998; SI Units for Clinical Measurement; American

College of Physicians; Philadelphia and Burtis, C.A, Ashwood, E.R and Bruns, D.E; 2008;

Fundamentals of Clinical Chemistry; Saunders Elsevier; Missouri [Laboratory test converted to

SI will be stored in SDTM LB domain as LBSTRESU and LBSTRESC]. Additionally, clinical

laboratory test results will be converted in Conventional Units, and store in SDTM SUPPLB

domain.

All clinical laboratory test results will be graded per NCI CTCAE v4.03 if applicable, as well as

high (higher than the normal range), normal (in the normal range) and low (lower than normal

range).

Descriptive statistics (n, mean, standard deviation, median, and range) of the lab parameters and

changes from baseline will be presented by regimen and dose group for biochemistry, hematology,

and coagulation. Such descriptive statistics will be presented at Baseline and at End of Study, as

well, Worst Result post Baseline (i.e. Maximum and Minimum post Baseline including results

from unscheduled assessments) will be presented as well.

Shift in biochemistry, hematology, and coagulation result CTCAE grading from baseline will be

tabulated at the end of treatment, as well as from baseline to the maximal grade during the study

(maximal grade will also include results from unscheduled and repeated assessments).


Related to: SOP-GDO-WW-019

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

All clinical laboratory test results will be listed in the original, SI, and Conventional units, for

biochemistry, hematology, coagulation, and urinalysis.

Individual patient biochemistry, hematology, and coagulation parameters during the trial can be

presented graphically using longitudinal spaghetti plots. Specific lab parameters to be plotted will

be decided by Symphogen from clinical meaning perspective after examination of corresponding

listings.

Biochemistry, hematology, and coagulation parameters will be presented using box plots by visits

and tumor type.

Results from the pregnancy tests will be listed.

4.11.5 Electrocardiogram

ECG parameter data will be listed by part dose group, time point, and patient.

Normal, abnormal, or abnormal clinically significant ECG will be summarized by regimen, dose

at Baseline, EOT and Worst Post Baseline; as well, a shift table from baseline to EOT and Worst

Post Baseline will be summarized by cohort. Number and percentage of patients with end of

treatment and maximum postdose QTcF values of <=450, >450 ms and <=480, >480 ms and

<=500, and >500 ms, and maximal change from baseline values of <=30, >30 <=60ms, and >60

ms will be summarized by part and dose group (highest QTcF Prolongations measurement will

also include results from unscheduled assessments). Above categories of QTcF are based on ICH

E14[2].

4.11.6 Echocardiogram (ECHO) or Multi-Gated (MUGA) Scan

ECHO/MUGA data will be listed.

4.11.7 Vital Signs and Body Measurements

Data for vital signs (body weight, blood pressure, heart rate, temperature) will be listed by part,


dose group, patient, at Baseline and EOT.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

Descriptive summary statistics (for observed values and changes from baseline) for vital sign

parameters (blood pressure and heart rate) will be provided for Baseline, EOT and Worst Result

post Baseline (i.e. Maximum and Minimum post Baseline including results from unscheduled

assessments) by regimen and dose group.

4.11.8 Physical Examination

All abnormal findings from the physical exam will be listed.

A shift table from baseline to EOT and worst from baseline of normal and abnormal findings in

physical examination by regimen and cohort will be produced.

4.11.9 Eastern Cooperative of Oncology Group (ECOG) Performance Status (PS)

ECOG performance status will be listed and summarized by shift table from baseline to EOT and

worst from baseline.

4.11.10Safety Monitoring (Independent Data Monitoring Committee [IDMC], Data

Monitoring Committee [DMC], Data and Safety Monitoring Board [DSMB])

A safety monitoring committee (SMC) was be established and included Investigator(s), Medical

Monitor(s) and Sponsor's medical representatives. The SMC reviewed clinical and laboratory

safety data regularly throughout the trial and will select the RP2D and regimen to be used in Part

2 based on safety data, as well as available PK and target engagement results. Additionally, the

annual Development Safety Update Report (DSUR) was submitted by Symphogen or designee to

all appropriate HAs and central IRBs/ECs as per ICH Guidelines. Submission of the DSUR to

local IRBs/ECs has been handled as per local regulations and/or requests.

4.12 Other Analyses

No other analyses.

4.13 Determination of Sample Size

No formal testing of hypotheses has been planned in this study. Therefore, no formal sample size

calculations were performed.

Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

4.14 Changes in the Conduct of the Study or Planned Analysis

The trial has been stopped during Part 1, no patient is enrolled in Part 2. Part 2 of the trial did not

take place.

• Objectives for Part 2 are omitted. Per protocol, the concentration of total Pan-HER (the

sum of the serum concentration for all six mAbs) was planned to be used for the PK

analysis. However, in an exploratory analysis, the PK of the six mAbs was shown not to

be similar, and hence using the sum of concentrations is not justified. Hence, the PK of

each mAb is reported;

• Overall Survival was planned as one of the Protocol Endpoints, this analysis will not be

performed: patients in this study are not followed up to death so that OS would resulted in

a truncated biased estimate;

• Time to documented PD, death, patient withdrawal or end of trial participation, whichever

comes first was initially planned in the Protocol Endpoints. Actually, based on FDA

guideline as of December 2018 [3], TTP is mentioned as a possible endpoint for

oncological studies, 'TTP is defined as the time from randomization until objective tumor

progression; TTP does not include deaths.'. TTP will be used an endpoint in this study

instead of the planned time to documented PD, death, patient withdrawal or end of trial

participation.

• Duration of SD was initially planned in the Protocol Endpoints, anyway this endpoint is

overlapping with TTP being derived in a very similar way; thus, this endpoint will not be

part of the data analysis.

DCR analysis was not included as part of study endpoints in the Protocol, such analysis

has been added in this SAP.

Given the early interruption of the trial, Symphogen decided to proceed with an abbreviated

Clinical Study Report; from list of Tables, Figures and Listings reported in below section 6, only

those flagged with asterisk (\*) will be produced for the abbreviated CSR.


Related to: SOP-GDO-WW-019


Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

## 5 REFERENCES

- [1] E.A. Eisenhauer et Al. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). EUROPEAN JOURNAL OF CANCER2009; 45;228-247.
- [2] ICH HARMONISED TRIPARTITE GUIDELINE; THE CLINICAL EVALUATION OF QT/QTC INTERVAL PROLONGATION AND PROARRHYTHMIC POTENTIAL FOR NON-ANTIARRHYTHMIC DRUGS; E14.
- [3] Clinical Trial Endpoints for the Approval of Cancer Drugs and Biologics, December 2018, U.S. Department of Health and Human Services Food and Drug Administration Oncology Center of Excellence.
- [4] SAS® Version 9.3. SAS Institute Inc. SAS and all other SAS Institute Inc. product or service names are registered trademarks or trademarks of SAS Institute Inc., Cary, NC, USA.

# Statistical Analysis Plan Template for Early Phase Studies

Symphogen A/S Sym013-01

# 6 TABLES, FIGURES AND LISTINGS

All the Tables, Figures and Listings with asterisk will be included in the CSR.

- Table 14.1.1 Patient Enrollment (All Consented Patients) \*
- Table 14.1.2 Patient Disposition by Treatment Schedule and Dose Group (Full Analysis Set) \*
- Table 14.1.3 Patient Demographics and Baseline Characteristics (Full Analysis Set) \*
- Table 14.1.4 Cancer Baseline Characteristics (Full Analysis Set)
- Table 14.1.5 Prior Cancer Therapies (Full Analysis Set)
- Table 14.2.1.1 Serum Concentration of the six monoclonal antibodies in Pan-HER for single and repeated dose PK profiles (Full Analysis Set) \*
- Table 14.2.1.2 Peak and Trough Serum Concentration of the six monoclonal antibodies in Pan-HER by Study Day (Full Analysis Set) \*
- Table 14.2.2 Serum PK Parameters for the six monoclonal antibodies in Pan-HER (Full Analysis Set) \*
- Table 14.2.3.1 Biomarkers from Skin Biopsy (Full Analysis Set) \*
- Table 14.2.3.2 Biomarkers from Tumor Biopsy (Full Analysis Set) \*
- Table 14.2.4.1 Best Overall Response Objective Response and Disease Control Rate (Full Analysis Set) \*
- Table 14.2.4.2 Time to Progression (Full Analysis Set) \*
- Table 14.2.4.3 Maximal Reduction in Sum of Diameters of Target Lesion from Baseline (Full Analysis Set)
- Table 14.2.4.4 Maximal Reduction in Sum of Diameters of Target Lesion from Baseline by Primary Tumor Type (Full Analysis Set)


Table 14.2.4.5 Number of Treatment Cycles (Full Analysis Set) \*


Symphogen A/S Sym013-01

Table 14.2.4.6 Treatment Duration and Dose Intensity (Full Analysis Set) \*

Table 14.2.4.7 Dose Reduction, Interruption, and Delay (Full Analysis Set) \*

Table 14.2.4.8 Dose-Limiting Toxicity (DLT Set) \*

Table 14.3.1.1 Overall Summary of TEAEs (Full Analysis Set) \*

Table 14.3.1.2 TEAEs by SOC and PT (Full Analysis Set) \*

Table 14.3.1.3 Related TEAEs by SOC and PT (Full Analysis Set) \*

Table 14.3.1.4 TEAEs by SOC and PT and Worst CTCAE Grade (Full Analysis Set) \*

Table 14.3.1.5 Related TEAEs by SOC and PT and Worst CTCAE Grade (Full Analysis Set) \*

Table 14.3.1.6 Serious TEAEs by SOC and PT (Full Analysis Set) \*

Table 14.3.1.7 Related Serious TEAEs by SOC and PT (Full Analysis Set) \*

Table 14.3.1.8 TEAEs Leading to Permanent Discontinuation of IMP by SOC and PT (Full Analysis Set) \*

Table 14.3.1.9 Related TEAEs Leading to Permanent Discontinuation of IMP by SOC and PT (Full Analysis Set) \*

Listing 14.3.2.1 Serious Adverse Events - Key Patient Information (Full Analysis Set) \*

Listing 14.3.2.2 Adverse Events with Outcome of Death - Key Patient Information Full Analysis Set \*

Listing 14.3.2.3 Adverse Events Leading to Permanent Discontinuation of Investigational Product - Key Patient Information Full Analysis Set \*

Listing 14.3.2.4 Adverse Events Leading to Dose Reduction - Key Patient Information Full Analysis Set \*

Listing 14.3.2.5 Adverse Events Leading to Infusion Interruption or Stop - Key Patient Information Full Analysis Set \*


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

Symphogen A/S Sym013-01

Listing 14.3.2.6 Listing of Death- Key Patient Information (Full Analysis Set) \*

Listing 14.3.4.1 Abnormal Hematology Values \*

Listing 14.3.4.2 Abnormal Chemistry and Coagulation Values \*

Listing 14.3.4.3 Abnormal Urinalysis Values \*

Table 14.3.5.1 Clinical Laboratory Hematology-Summary of Observed Values and Change from Baseline (Full Analysis Set) \*

Table 14.3.5.2 Clinical Laboratory Chemistry-Summary of Observed Values and Change from Baseline (Full Analysis Set) \*

Table 14.3.5.3 Clinical Laboratory Coagulation-Summary of Observed Values and Change from Baseline (Full Analysis Set) \*

Table 14.3.5.4 Clinical Laboratory Hematology -Summary of CTCAE Grade Shift from Baseline to Maximal Grade (Full Analysis Set) \*

Table 14.3.5.5 Clinical Laboratory Chemistry –Summary of CTCAE Grade Shift from Baseline to Maximal Grade (Full Analysis Set) \*

Table 14.3.5.6 Clinical Laboratory Coagulation –Summary of CTCAE Grade Shift from Baseline to Maximal Grade (Full Analysis Set) \*

Table 14.3.6.1 Vital Signs and Weight Observed Values and Change from Baseline (Full Analysis Set) \*

Table 14.3.6.2 ECG Clinical Assessment (Full Analysis Set) \*

Table 14.3.6.3 ECG Shift from Baseline (Full Analysis Set) \*

Table 14.3.6.4 ECG- QTcF Prolongations Summary (Full Analysis Set) \*

Table 14.3.6.5 Physical Examination Clinical Assessment (Full Analysis Set)

Table 14.3.6.6 Physical Examination Shift from Baseline (Full Analysis Set) \*

TP-GDO-WW-133-01 CONFIDENTIAL Project Document Version No. Final 1.0 Effective Date: 05 Sep 18 Project Document Effective Date: 05 April 2019 Related to: SOP-GDO-WW-019 

Symphogen A/S Sym013-01

Table 14.3.6.7 ECOG-PS (Full Analysis Set)

Table 14.3.6.8 ECOG-PS Shift from Baseline (Full Analysis Set) \*

Figure 14.2.1 Skin Biopsy: scatter plot of EGFR receptors down modulation at C1D8 and C1D15 versus Baseline (Full Analysis Set) \*

Figure 14.2.2 Skin Biopsy: scatter plot of HER3 receptors down modulation at C1D8 and C1D15 versus Baseline (Full Analysis Set) \*

Figure 14.2.3 Skin Biopsy: scatter plot of Ki67 receptors down modulation at C1D8 and C1D15 versus Baseline (Full Analysis Set) \*

Figure 14.2.4 Tumor Biopsy: scatter plot of EGFR receptors down modulation at End of Cycle 2 versus Baseline (Full Analysis Set) \*

Figure 14.2.5 Tumor Biopsy: scatter plot of HER2 receptors down modulation at End of Cycle 2 versus Baseline (Full Analysis Set) \*

Figure 14.2.6 Tumor Biopsy: scatter plot of HER3 receptors down modulation at End of Cycle 2 versus Baseline (Full Analysis Set) \*

Figure 14.2.7 Tumor Biopsy: scatter plot of Ki67 receptors down modulation at End of Cycle 2 versus Baseline (Full Analysis Set) \*

Figure 14.2.8 Pharmacokinetics of PanHer Monoclonal Antibodies: Patient Profiles for concentration versus actual time by Monoclonal Antibody, Dose Schedule and Dose Group (First and Second Profiles) – Linear (Full Analysis Set) \*

Figure 14.2.9 Pharmacokinetics of PanHer Monoclonal Antibodies: Patient Profiles for concentration versus actual time by Monoclonal Antibody, Dose Schedule and Dose Group (First and Second Profiles) – Semi-Log (Full Analysis Set) \*

Figure 14.2.10 Pharmacokinetics of PanHer Monoclonal Antibodies: Single Patient Profiles for concentration versus actual time (all Monoclonal Antibodies overlaid) (First and Second Profiles) – Semi-Log (Full Analysis Set) \*


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 Project Document Version No. Final 1.0 Project Document Effective Date: 05 April 2019 

Symphogen A/S Sym013-01

Figure 14.2.11 Pharmacokinetics of PanHer Monoclonal Antibodies: Patient Profiles for concentration versus actual time by Monoclonal Antibody, Dose Schedule and Dose Group (peak and trough for each dosing occasion) – Linear (Full Analysis Set) \*

Figure 14.2.12 Pharmacokinetics of PanHer Monoclonal Antibodies: Patient Profiles for concentration versus actual time by Monoclonal Antibody, Dose Schedule and Dose Group (peak and trough for each dosing occasion) – Semi-Log (Full Analysis Set) \*

Figure 14.2.13 Pharmacokinetics of PanHer Monoclonal Antibodies: Single Patient Profiles for concentration versus actual time (all Monoclonal Antibodies overlaid) (peak and trough for each dosing occasion) – Semi-Log (Full Analysis Set) \*

Figure 14.2.14 Arithmetic Mean Concentration vs. planned time for each of the six mAbs by Dose Group (First and 2nd profiles) – Linear (Full Analysis Set) \*

Figure 14.2.15 Geometric Mean Concentration vs. planned time for each of the six mAbs by Dose Group (First and 2nd profiles) – Semi-Log (Full Analysis Set) \*

Figure 14.2.16 Arithmetic Mean Peak and Trough Concentrations for each of the six mAbs versus planned time point by Dose Group (peaks and troughs at all dosing occasions) – Linear (Full Analysis Set) \*

Figure 14.2.17 Geometric Mean Peak and Trough Concentrations for each of the six mAbs versus planned time point by Dose Group (peaks and troughs at all dosing occasions) – Semi-Log (Full Analysis Set) \*

Figure 14.2.18 Spaghetti Plot for Selected Hematology parameters (Full Analysis Set) \*

Figure 14.2.19 Spaghetti Plot for Selected Biochemistry parameters (Full Analysis Set) \*

Figure 14.2.20 Spaghetti Plot for Selected Coagulation parameters (Full Analysis Set) \*

Figure 14.2.21 BoxPlot for Selected Hematology parameters by Visit (Full Analysis Set)

Figure 14.2.22 BoxPlot Plot for Selected Biochemistry parameters by Visit (Full Analysis Set)

Figure 14.2.23 BoxPlot Plot for Selected Coagulation parameters by Visit (Full Analysis Set)


Symphogen A/S Sym013-01

- Figure 14.2.24 BoxPlot for Selected Hematology parameters by Visit and Tumor Type (Full Analysis Set)
- Figure 14.2.25 BoxPlot Plot for Selected Biochemistry parameters by Visit and Tumor Type (Full Analysis Set)
- Figure 14.2.26 BoxPlot Plot for Selected Coagulation parameters by Visit and Tumor Type (Full Analysis Set)
- Figure 14.2.27 Waterfall Plot of the Best Percent Change from Baseline in Sum of Diameters of Target Lesions (Full Analysis Set) \*
- Figure 14.2.28 Waterfall Plot of the Best Percent Change from Baseline in Sum of Diameters of Target Lesions by Primary Tumor Type (Full Analysis Set) \*
- Figure 14.2.29 Kaplan Meier Survival Curve for Time To Progression (Full Analysis Set) \*
- Figure 14.2.30 Swimmer Plot of Duration of Treatment and Tumor Response (Full Analysis Set)
  \*
- Listing 16.2.1.1 Patients Disposition (All Consented Patients) \*
- Listing 16.2.1.2 Screen Failure and Patients Not Meeting Eligibility Criteria (All Consented Patients) \*
- Listing 16.2.2.1 Protocol Deviations and Violations (All Consented Patients) \*
- Listing 16.2.3.1 Analysis Sets (All Consented Patients) \*
- Listing 16.2.4.1 Demographics and Baseline Characteristics (All Consented Patients) \*
- Listing 16.2.4.2 Medical and Surgical History (All Consented Patients) \*
- Listing 16.2.4.3.1 Prior and Concomitant Medications (All Consented Patients) \*
- Listing 16.2.4.3.2 Prophylactic Pre-medications (All Consented Patients) \*
- Listing 16.2.4.3.3 Concomitant Procedures (All Consented Patients) \*

TP-GDO-WW-133-01 CONFIDENTIAL Project Document Version No. Final 1.0
Effective Date: 05 Sep 18
Related to: SOP-GDO-WW-019


Symphogen A/S Sym013-01

Listing 16.2.4.4.1 Cancer Diagnosis (All Consented Patients) \*

Listing 16.2.4.4.2 Cancer Gene Mutation (All Consented Patients) \*

Listing 16.2.4.4.3 Prior Cancer Therapies: Surgical Procedure (All Consented Patients) \*

Listing 16.2.4.4.4 Prior Cancer Therapies: Radiation Therapy (All Consented Patients) \*

Listing 16.2.4.4.5 Prior Cancer Therapies: Systemic Therapy (All Consented Patients) \*

Listing 16.2.4.4.6 Prior Anti-EGFR Anti-HER2 Therapies (All Consented Patients) \*

Listing 16.2.5.1 Study Drug Administration (Full Analysis Set) \*

Listing 16.2.5.2 Study Drug Administration Irregularities (Full Analysis Set) \*

Listing 16.2.5.3 Study Drug Infusion Related Reaction (Full Analysis Set) \*

Listing 16.2.6.1 Pharmacokinetic Blood Sampling and Serum Concentrations of the six monoclonal antibodies in Pan-HER (Full Analysis Set) \*

Listing 16.2.6.2 Serum PK Parameters for the six monoclonal antibodies in Pan-HER (Full Analysis Set) \*

Listing 16.2.6.3 Pharmacodynamics Parameters, Biomarkers from Blood and Anti-Drug Antibody (Full Analysis Set) \*

Listing 16.2.6.4 Biomarkers from Skin Biopsy (Full Analysis Set) \*

Listing 16.2.6.5 Biomarkers from Archival Tumor/Tumor Biopsy (Full Analysis Set) \*

Listing 16.2.6.6 Tumor Markers (Full Analysis Set) \*

Listing 16.2.6.7.1 Tumor Assessment - Target Lesion (Full Analysis Set) \*

Listing 16.2.6.7.2 Tumor Assessment – Non-Target Lesion (Full Analysis Set) \*


Listing 16.2.6.7.3 Tumor Response by Visit (Full Analysis Set) \*

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 Project Document Version No. Final 1.0
Project Document Effective Date: 05 April 2019


Symphogen A/S Sym013-01

Listing 16.2.6.7.4 Best Overall Response, Objective Response, Time To Progression, Disease Control Rate (Full Analysis Set) \*

Listing 16.2.7.1 Dose Limiting Toxicity (DLT Analysis Set) \*

Listing 16.2.7.2.1 Adverse Events (All Consented Patients) \*

Listing 16.2.8.1 Clinical Laboratory Hematology Results and Change from Baseline (All Consented Patients) \*

Listing 16.2.8.2 Clinical Laboratory Chemistry and Coagulation Results and Change from Baseline (All Consented Patients) \*

Listing 16.2.8.3 Clinical Laboratory Urinalysis Results (All Consented Patients) \*

Listing 16.2.8.4 Pregnancy Test (All Consented Patients) \*

Listing 16.2.9.1 Vital Signs – Observed and Change from Baseline Values (All Consented Patients) \*

Listing 16.2.9.2 Electrocardiogram (All Consented Patients) \*

Listing 16.2.9.3 ECHO/MUGA(ECHO) (All Consented Patients) \*

Listing 16.2.9.4 Physical Examination (All Consented Patients)

Listing 16.2.9.5 ECOG-PS (All Consented Patients) \*

TP-GDO-WW-133-01 CONFIDENTIAL Project Document Version No. Final 1.0 Effective Date: 05 Sep 18 Project Document Effective Date: 05 April 2019 Related to: SOP-GDO-WW-019 

Symphogen A/S Sym013-01

# 7 APPENDICES

# 7.1 Schedule of Assessments Q1W dosing

| Pre-Treatment Period | | | | | | | | Treatm | Freatment Period | , pos | | | | | | Post-Treatu | Post-Treatment Period |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | Cycle 1 | | | | Č | Cycle 2, 4, 6 etc | 6 etc. | | | Crde 3, | . S. 7 etc | | EOT | IM FUP |
| Day within Cycle<br>Visit Window (= days) | D-14 to<br>D-1 | īQ | 8 | ST. | <u>23</u> | 87 | E 2 | 83 | 51G | HI | End of<br>Cycle | a? | 80 <del>⊕</del> | 10.05 | 87 | 2 10 d from the decision of that treatment | I mouth after<br>last dose of trial<br>treatment |
| Informed Cousent | X | 1 | | | | | | | | | | | | | | TO ALCOHOLD THE PARTY OF THE PA | 1 |
| Baseline Charactensucs*Eligibility | X | X | | | | | | | | | | | | | | | |
| Safety Assessments | | | | | | | | | | | | | | | - | | |
| Medication Procedure Survey | X | X | N. N. | × | X | X | × | × | × | × | X | X | × | × | X | ** | × |
| (S)AE Survey and Reporting | X | (X) | (X) | × | X | X | X | X | X | X | (X) | X | X | X | × | X | X |
| DLT Evaluation* Part I only | | (X) | X | × | × | X | Class vilus | | | | | | | | | | |
| ital Signs and Body Measurements | X | X | | × | X | X | × | × | × | × | | X | X | X | × | X | X |
| ECO 6 PS | X | X | | | | | × | | | | | X | | | | X | X |
| Physical Evanzination | X | N. | | | | | × | | | | | × | | | | X | X |
| ECG. | X | | | | | | 300 | | | | | | | | | (X) | |
| ECHO or MUGA scan | X | | 3 | | 3 | Sec. 1 | 1 | | | | | - | | The same of | | X | |
| Safety blood samples "" | X | | X | × | × | X | N | | × | | | X | | X | | X | X |
| Trinalysis <sup>6,8</sup> | X | N. | | | X | 0 | × | | 120 | | 120 | X | | | | X | X. |
| Pregnancy Test | X | | | | | | | | | | | | | | | N. | |
| Complement Panel <sup>10</sup> Part 2 only | | X | 7 | | 200 | Ì | | | | | | | | | | The second second | |
| Disease Assertments | - 201 | | 70 | | - | | | | | | 2 | | - 25 | - 15 | - 15 | 100 | |
| | X | | | | | | | | | | EX. | | | | | XII | XII |
| Tumor Marker Evaluation, if applicable " | X | | 100 | | | | The state of the s | | 100 | | No. | | | | | N | X |
| Archival Tumor Tissue" Part 1: Submit if available (optional) | х | | | | | | | | | | | | | | | | |
| Additional Assessments | 200 | Same? | of Second | 1 | Sec. 125 | Section of the last | 100 | Section 1 | 100 | | ( ) | S 1000 | The second | | 1000 | 2007 (3) | 2000 |
| PK Samples ** | | ** | (X) | × | × | X | × | X | X | × | | X | × | X | X | X | X |
| ADA Sample | | X | | | | | ខង្ខ | | | | | 8 | | | | X | X |
| Skin Biopsy <sup>16</sup> | X | | | × | X | | | | | | | | | | | | |
| Tumot Biopsy <sup>17</sup> Part 1: Optional Part 2: Required | X | | | | | | | | | | C) only | | | | | | |
| Biomarker Blood Sample 18 | X | | | | | | | | | | C2 only | | | | | X | 144 |
| rial Treatment | | | | | | | | | | | | | | | | | |
| Pan-HER Premedication" | | X | | × | × | X | × | × | × | × | -0 | X | × | × | × | | |
| an-HER Infusion | | X | | × | X | X | × | × | X | × | | 1 | × | X | X | | |

Abbreviations (in alphabetical order). ADA, anni-drug antibody. C. Cycle; CT, computed tomography. Did. day(s); DLT, dose-limiting toxicity; EOT, End of Treatment: ECG, electrocardiogram; ECOG PS, Eastern Cooperative Oncology Group performance stems; MRI, magnetic resonance imaging, MUGA, multi-gated acquisition; IM FUP, 1-Month Follow-up, PK, pharmacokimetic; (5)AE, (serious) adverse event

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

CONFIDENTIAL Project Document Version No. Final 1.0

Project Document Effective Date: 05 April 2019


# Statistical Analysis Plan Template for Early Phase Studies PAREXEL International

Symphogen A/S Sym013-01

- The treatment period courtaines until the patient is withdrawn from Pan-HER.
- Survival follow-up is required until death, withdrawal of consent, or termination of the trial. This continued follow-up does not require an in-person visit at the trial site, but mouths. Response assessment follow-up is required in the event of an ongoing SD, PR or CR at the 1M FUP Visit, until PD or another therapeutic intervention is initiated Applicable for Part 2 only: After the 1M FUP Visit, the Investigator will make every effort to obtain follow-up information on response assessment and or OS every 2 may be obtained by collection of data documentation
- Informed consent may be obtained outside the 14-day screening period prior to C.I.D., but is recommended to be obtained no earlier than 4 weeks prior to the planned C.I.D.1
- Screening assessments baseline characteristics include demographics, medical history, nunor histology, mutation status, extent of disease, prior auti-caucer peatment etc.
  - DLT evaluation, Applicable for Part 1 only: DLTs are reported during Cycle 1 with final assessment 7 days after the last dose of Cycle 1 or prior to dosing on C2 D1.
- Does not need to be performed on CLD1 if performed during screening 2.7 days from CLD1.
- In addition to the scheduled tunepoints, an ECG should be performed in the event of cardiac symptoms.
- In addition to the scheduled timepoints, an ECHO MUGA should be performed in the event of cardiac symptoms
- Local laboratory results must be available and assessed prior to each Pan-HER infusion for all ministons during Cycle 1, and for every second infusion from Cycle 2 ouwards. Refer to Section 8.2.9 for further details
- Complement sampling. Applicable for Part 2 only, will be done C1D1 and in the event of an IRR. Refer to Section \$2.10 for further details Complement sampling, Applicable for Part 2 only, will be done CL.
   CT or MFI unaging schedule and conditions, applying to all cohorts.
- A CTARI performed within 18 days prior to CLD1 can be used for evaluation of eligibility and as baseline scan, provided that the CTARI has been performed according to the clinical trial protocol requirements
- The first CTMRI assessment for response is done at the end of Cycle 2 and thereofter repeated at the end of every second cycle (in the week prior to Day 1 of the next
- In the event of suspected PD, a CT MRI is to be performed as soon as possible.
- In the event of CR.PR, a confirmatory CT.MRI is to be performed 28 (+7) days after the first assessment of CR.PR.
- 12) A CTMRI at EOT should only be performed if the previous CTMRI has been performed 3 weeks before, a CTMRI scan at 1M FUP aboutd only be performed if no CT MRI documents disease progression before or at EOT
- 13) Tumor marker evaluation to include tumor markers that are part of the trial site standard practices as inducated by rumor type, if applicable
- 14) Archival tumor fissue, applicable for patients in Part 1 only if tissue is available. To be assessed locally, preferably by immunohistochemistry (HC). Does not need to be repeased if EGFR and HER2 status have been assessed previously and the pathology report is available to document findings
- Extended PK sampling for PK profiling will be done starting Cl.Dl and Cl.Dll. Refer to Table 11 for further details.
- 16) Skin biopsy. All panents earolled will undergo skin biopsies. Sample is to be obtained during screening after patient eligibility has been confirmed. Sampling is to be repeated Cycle 1 Day 8 (prior to dosing) and Cycle 1 Day 15 (prior to dosing).
  - 17) Tumor biopsy, Optional for patients in Part 1. Required for all patients in Part 2: To be assessed centrally. Tumor biopsy is to be performed after patient eligibility has been confirmed. Archival dismanne and proceed at screening if suitable for central analysis. Sampling is repeated at the end of Cycle 2 or upon PD, whichever occurs first Refer to Section 8.7 for further details
- 18) Biomarker blood sample. To be obtained during screening after patient eligibility has been confinmed. Sampling is to be repeated at the end of Cycle 2 or upon PD, whichever occurs first, and at EOT
  - 19) Premedication. For Part 1, premedication is mandatory prior to each dose of Pan-HER. For Part 2, premedication is mandatory prior to each dose of Pan-HER during Cycle 1. In Par 2, premedication may be withdrawn after Cycle 2 on a patient-by-panent basis, if the patient is without evidence of IRRs. Refer to Section 7.2.1 for details


# Statistical Analysis Plan Template for Early Phase Studies PAREXEL International

Symphogen A/S

# Symo13-01 7.2 Schedule of Assessments Q2W dosing

| Pre-Treatment Period | | | | | | | Treatment Period | r Period | | | | Post-Treats | Post-Treatment Period <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | ľ | Cycle.1 | | T | 0 | Cycle 2, 4, | 6 etc. | Cycle 3. | 1. 5. 7 etc. | EOT | 1M FUP |
| Day within Cycle<br>Visit Window (= days) | D-14 to | 8 | 60 | D8 (=2) | 12 G | EG. | E T | E | End of Cycle | Ea | SIG. | ≤ 10 d from the decision of trial treatment withdrawal | I month after<br>last dose of trial<br>treatment<br>(30-74) |
| Informed Consent | X | | | | | 100 | | | | 200 | | The state of the s | The second second |
| Baseline Characteristics / Eligibility | (X) | EX. | | | | | | | | | | | |
| Safety Assessments | | The second | Section 1 | 1 | 3 | Section 1 | - | The second | | 1000 | 1 | *** | 100 |
| Medication Procedure Survey | × | No. | N.X. | × | X | X | × | X | X | × | X | X | X |
| 5) AE Survey and Reporting | X | OX S | X | × | X | X | × | X | X | | (X) | X | X |
| DLT Evaluation Part I only | | X | X | X | X | X | C2 only | - | 1000 | 200 | | | |
| Vital Signs and Body Measurements | (X) | N. | | X | (X) | X | X | (X) | | X | X | X | X |
| ECOG PS: | X | X | | | - | | × | | | X | | X | X |
| Physical Evanumation: | X | X | | | | | × | | | × | | X | X |
| :508 | X | | | | | | | | | | | X | |
| ECHO or MUGA scans | × | 1 | Sec. and | 1000 | 10.00 | 1 | 1000 | · Alexandra | | 2000 | | X | 1000 |
| Safety blood samples "" | X | X | X | X | X | X | X | X | | X | X | X | X |
| Urinalysis** | × | X | | | X | | × | | | X | | X | X |
| Pregnancy Test | X | | | | | | 100 | | | | | X | |
| Complement Panel " Part 2 only | | X | | | | | | | | | | | |
| Disease Assessments | 4000 | | | | | 200 | | | 2000 | N.C | | W | 100 |
| Disease Status Evaluation by CT/ MRI'!! | X X | | | | | | | | X | | | N <sub>15</sub> | XII |
| l'amor Marker Evaluation, if applicable | X | | 100 | | | | | | X | | 200 | X | X |
| Archival Tumor Tissue <sup>14</sup> Part I: Submit if available (optional) | х | | | | | | | | | | | | |
| Additional Assessments | | | Sec. 1 | 2 | | Sec. of | - | The second second | - | 10000 | The second | *** | |
| PK Samples ** | | X | N. X | X | X | X | X | X | | X | (X) | X | X |
| ADA Sample | | X | | | | | C3 only | | | X | | X | х |
| Skin Biopsy** | X | | 20 | × | X | 34 | | | No. | 332 | | | |
| Tumor Biopsy Part 2: Required | х | | | | | | | | CJ endy | | | | |
| Biomarker Blood Sample <sup>18</sup> | X | | | | | | | | C2 only | | | X | |
| Irial Treatment | | Į | | | | | | | | - | - | | |
| Pan-HER Premedication " | | N. | 9 | | X | 3 | X | X | | X | X | 9 | |
| Pan-HER Infusion | | X | | | X | 07 | × | X | | X | No. | | |
| Post-Infusion Monitoring | | (X) | | | X | | × | X | | X | X | ALC: NO PERSON NAMED IN COLUMN | |

Abbreviations (in alphabetical order): ADA, sun-drug antibody; C, Cycle; CT, computed tomography; D/d, day(s); DLT, dose-limiting toxicity; EOT. End of Treatment Visit: ECG, electrocardogram; ECHO, echocardiogram; ECHO,

Related to: SOP-GDÖ-WW-019 Effective Date: 05 Sep 18 TP-GDO-WW-133-01


 Project Document Version No. Final 1.0 Project Document Effective Date: 05 April 2019

# Symphogen A/S Sym013-01

- 1) The treatment period continues until the patient is withdrawn from Pan-HER
- Survival follow-up is required until death, withdrawal of consent, or termination of the trial. This couranted follow-up does not require an in-person visit at the trial site, but months. Response assessment follow-up is required in the event of an ongoing SD, PR or CR at the IM FUP Visit, until PD or another therapeutic intervention is immared Applicable for Part 2 only: After the LM FUP Visit, the Investigator will make every effort to obtain follow-up information on response assessment and or OS every 2 may be obtained by collection of data documentation
- Informed consent may be obtained outside the 14-day screening period prior to CLD1, but is recommended to be obtained no earlier than 4 weeks prior to the planned CLD1
  - Screening assessments baseline characteristics include demographics, medical history, rumor histology, mutation status, extent of disease, prior auti-caucer meatment arc.
    - DLT evaluation. Applicable for Part 1 only: DLTs are reported during Cycle 1 with final assessment 7 days after the last dose of Cycle 1 or prior to dosing on C2D1
- Does not need to be performed on C1D1 if performed during screening ≤ 7 days from C1D1.
- In addition to the scheduled tunepoints, an ECG should be performed in the event of cardiac symptoms
- In addition to the scheduled timepoints, an ECHO MUGA should be performed in the event of cardiac symptoms
- Local laboratory results must be available and assessed prior to each Pan-HER unfusion for all unfusions during Cycle I, and for every second infusion from Cycle I ouwards. Refer to Section 8.2.9 for further details
- 10) Complement sampling. Applicable for Part 2 only, will be done C1 D land in the event of an IRR. Refer to Section 8.2.10 for further details
  - 11) CT or MFI unaging schedule and conditions, applying to all cohoms.
- A CIMIN performed within 18 days prior to CLDI can be used for evaluation of eligibility and as baseline scan, provided that the CIMIN has been performed according to the clinical trial protocol requirements
- The first CTMRI assessment for response is done at the end of Cycle 2 and thereafter repeated at the end of every second cycle (in the week prior to Day 1 of the next
- In the event of suspected PD, a CTARL is to be performed as soon as possible
- In the event of CR PR, a confirmatory CT MR1 is to be performed 18 (+7) days after the first assessment of CR PR.
- 12) A CTMRI at EOT should only be performed if the previous CTMRI has been performed >3 weeks before; a CTMRI scan at IM FUP should only be performed if no CT.MRI documents disease progression before or at EOI
  - Tumor marker evaluation to include tumor markers that are part of the trial site standard practices as indicated by numor type, if applicable
- 14) Archival rumor fissue, applicable for patients in Part 1 only if fissue is available. To be assessed locally, preferably by immunolistochemistry (IHC). Does not need to be repeated if EGFR and HERD status have been assessed previously and the pathology report is available to document findings
  - 15) Extended PK sampling for PK profiling will be done starting C1 D1 and C2 D1. Refer to Table 11 for further details
- 16) Skin biopsy: All parieurs emolibed will undergo skin biopsies. Sample is to be obtained during screening after patient eligibility has been confirmed. Sampling is to be repeated Cycle 1 Day 8 and Cycle 1 Day 15 (prior to dosing)
- Tumor biopsy. Optional for patients in Part 1. Required for all patients in Part 2. To be assessed centrally Tumor biopsy is to be performed after patient eligibility has been confirmed. Archival itssue may be accepted at screening if suitable for central analysis. Sampling is repeated at the end of Cycle 2 or upon PD, whichever occurs first. Refer to Section 8.7 for further details E
- 13) Biomarker blood sample. To be obtained during screening after patient eligibility has been confirmed. Sampling is to be repeated at the end of Cycle 2 or upon PD, whichever occurs first, and at EOT. For those timepoints where both a blood sample and a tumor biopsy are to be obtained, blood sample to be collected first.
- prophylaxis is mandatory during Cycle 1 and Cycle 2. Thereafter, if the patient is without evidence of IRRs or mucositis, the Investigator may choose to withdraw related Premedication. For Part I, intensive prophylaxis, as defined berein, on a mandatory basis is required to reduce the risk of IRRs and oropharyngeal mucositis. For Part 2, medications with subsequent dosing. Refer to Sections 7.2.1 and 7.2.2 for details 61


Symphogen A/S Sym013-01

# 7.3 Derivation of CTCAE Grade - Hematological Tests

| Tests | Direction | | Gra | Grade | |
|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 |
| Hemoglobin (g/dl, | $\rightarrow$ | <lln -="" 10.0="" dl;<="" g="" td=""><td>&lt;10.0 - 8.0 g/dL;</td><td>&lt;8.0 g/dL;</td><td>Life-threatening</td></lln> | <10.0 - 8.0 g/dL; | <8.0 g/dL; | Life-threatening |
| mmol/L | | <lln -="" 6.2<="" td=""><td>&lt;6.2 - 4.9 mmol/L;</td><td>&lt;4.9 mmol/L;</td><td>conseduences;</td></lln> | <6.2 - 4.9 mmol/L; | <4.9 mmol/L; | conseduences; |
| or g/L) | | mmol/L; | <100 - 80g/L | <80 g/L; | ı |
| | | <lln -100="" g="" l<="" td=""><td>•</td><td>,</td><td></td></lln> | • | , | |
| Platelet (/mm3 or | $\rightarrow$ | - NTT> | <75,000 - | <50,000 - | <25,000/mm3; |
| (T) | | 75,000/mm3; | 50,000/mm3; <75.0 | 50,000/mm3; <75.0 25,000/mm3; <50.0 | <25.0 x 10e9 / L |
| | | <lln -="" 10e9<="" 75.0="" td="" x=""><td>-50.0 x 10e9 /L</td><td>- 25.0 x 10e9 /L</td><td></td></lln> | -50.0 x 10e9 /L | - 25.0 x 10e9 /L | |
| | | 7/ | | | |
| Neutrophils (/mm3 | $\rightarrow$ | <lln -="" 1500="" mm3;<="" td=""><td><lln -="" 1000="" 1500="" 500="" <1000="" <1500="" mm3;="" mm3;<="" td="" =""><td>&lt;1000 - 500/mm3;</td><td>&lt;500/mm3; &lt;0.5 x</td></lln></td></lln> | <lln -="" 1000="" 1500="" 500="" <1000="" <1500="" mm3;="" mm3;<="" td="" =""><td>&lt;1000 - 500/mm3;</td><td>&lt;500/mm3; &lt;0.5 x</td></lln> | <1000 - 500/mm3; | <500/mm3; <0.5 x |
| or /L) | | <lln -="" 1.0="" 1.5="" <1.5="" l="" l<="" td="" x109="" x10e9="" =""><td><math>&lt;1.5 - 1.0 \times 10e9 / L</math></td><td>&lt;1.0 - 0.5 x 10e9 / L</td><td>10e9 /L</td></lln> | $<1.5 - 1.0 \times 10e9 / L$ | <1.0 - 0.5 x 10e9 / L | 10e9 /L |
| Lymphocyte (/mm3 | $\rightarrow$ | <lln -="" 800="" mm3;<="" td=""><td>&lt;800 - 500/mm3;</td><td>&lt;500 - 200/mm3;</td><td>&lt;200/mm3;</td></lln> | <800 - 500/mm3; | <500 - 200/mm3; | <200/mm3; |
| or /L) | | <LLN - 0.8 x10e9 $ <$ 0.8 - 0.5 x10e9 /L | <0.8 - 0.5 x10e9 /L | <0.5 - 0.2 x 10e9 / L | <0.2 x 10e9 /L |
| | | /T | | | |
| Note: $10e9 = 10^9$ ; LL | N = Lower Limit of N | Note: 10e9 = 109; LLN = Lower Limit of Normal; ULN = Upper Limit of Normal | imit of Normal | | |

CONFIDENTIAL Project Do

Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

TP-GDO-WW-133-01

Project Document Version No. Final 1.0 Project Document Effective Date: 05 April 2019 

# Statistical Analysis Plan Template for Early Phase Studies PAREXEL International

# Symphogen A/S Sym013-01 7.4 Derivation of CTCAE Grade – Clinical Chemistry Tests

| Toete | Direction | | opean | مام | |
|---|---|---|---|---|---|
| | DIICCIIOII | , | | | , |
| | | 1 | 2 | 3 | 4 |
| Sodium (mmol/L) | $\rightarrow$ | <lln -="" 130<br="">mmol/L</lln> | - | <130 - 120 mmol/L | <120 mmol/L |
| Sodium (mmol/L) | <b>←</b> | 1 | 150 >150 - 155 mmol/L | >155 - 160 mmol/L | >160 mmol/L |
| Potassium (mmol/L) | $\rightarrow$ | <lln -="" 3.0="" l<="" mmol="" td=""><td>1</td><td>&lt;3.0 - 2.5 mmol/L</td><td>&lt;2.5 mmol/L</td></lln> | 1 | <3.0 - 2.5 mmol/L | <2.5 mmol/L |
| Potassium (mmol/L) | <b>←</b> | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >5.5 - 6.0 mmol/L | >7.0 mmol/L |
| Glucose | $\rightarrow$ | <pre><lln -="" 55="" dl;<="" mg="" pre=""></lln></pre> <lln -="" 3.0="" l<="" mmol="" pre=""></lln> | <55 - 40 mg/dL;<br><3.0 - 2.2 mmol/L | <40 - 30 mg/dL;<br><2.2 - 1.7 mmol/L | <30 mg/dL;<br><1.7 mmol/L |
| Glucose | <b>←</b> | Fasting glucose value >ULN - | Fasting glucose value >160 - | >250 - 500 mg/dL;<br>>13.9 - 27.8mmol/L | >500 mg/dL;<br>>27.8 mmol/L |
| | | Fasting glucose value >ULN - 8.9 mmol/L | Fasting glucose value >8.9 - 13.9 mmol/L | | |
| Creatinine | ← | >1 - 1.5 x baseline;<br>>ULN - 1.5 x ULN | >1.5 - 3.0 x<br>baseline;<br>>1.5 - 3.0 x ULN | >3.0 baseline;<br>>3.0 - 6.0 x ULN | >6.0 x ULN |
| Bilirubin | ← | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN |
| Alkaline phosphatase (AKP) | - ← | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| AST (SGOT) | ← | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| ALT (SGPT) | ← | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Uric Acid | ↓ | >ULN - 10 mg/dL<br>(0.59 mmol/L) | 1 | 1 | >10 mg/dL;<br>>0.59 mmol/L |
| Calcium | <b>←</b> | Corrected serum | Corrected serum | Corrected serum | Corrected serum |

 Project Document Effective Date: 05 April 2019 Project Document Version No. Final 1.0 CONFIDENTIAL

Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

TP-GDO-WW-133-01

Symphogen A/S Sym013-01

| Tests | Direction | | Grade | ıde | |
|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 |
| | | calcium of | calcium of | calcium of | calcium of |
| | | Hypercalcemia | >11.5 - 12.5 mg/dL; | >12.5 - 13.5 mg/dL; | >13.5 mg/dL; |
| | | >ULN - 11.5 | 11.5 >2.9 - 3.1mmol/L; | >3.1 - 3.4 mmol/L; | >3.4 mmol/L; |
| | | mg/dL; | Ionized calcium | Ionized calcium | Ionized calcium |
| | | >ULN - 2.9 | >1.5 -1.6 mmol/L | >1.6 - 1.8 mmol/L | >1.8 mmol/L |
| | | mmol/L; | | | |
| | | Ionized calcium | | | |
| | | >ULN - 1.5 mmol/L | | | |
| Calcium | <b></b> | Corrected serum | Corrected serum | Corrected serum | Corrected serum |
| | | calcium of | calcium of | calcium of | calcium of |
| | | <LLN - 8.0 mg/dL; | <8.0 - 7.0 mg/dL; | < 8.0 - 7.0 mg/dL; | <6.0 mg/dL; |
| | | <lln -="" 2.0<="" td=""><td>&lt;2.0 - 1.75 mmol/L;</td><td>&lt;2.0 - 1.75 mmol/L;</td><td>&lt;1.5 mmol/L;</td></lln> | <2.0 - 1.75 mmol/L; | <2.0 - 1.75 mmol/L; | <1.5 mmol/L; |
| | | mmol/L; | Ionized calcium | Ionized calcium | Ionized calcium |
| | | Ionized calcium | <1.0 - 0.9 mmol/L; | <1.0 - 0.9 mmol/L; | <0.8 mmol/L; |
| | | <lln< td=""><td></td><td></td><td></td></lln<> | | | |
| | | -1.0 mmol/L | | | |
| Phosphate | <b>^</b> | <lln -="" 2.5="" <math="" dl;="" mg=""> &lt;2.5 - 2.0 mg/dL;</lln> | <2.5 - 2.0 mg/dL; | <2.0 - 1.0 mg/dL; | <1.0 mg/dL; |
| | | <lln -="" 0.6="" 0.8="" <0.8="" l="" l<="" mmol="" td="" =""><td>&lt;0.8 - 0.6 mmol/L</td><td>&lt;0.6 - 0.3 mmol/L</td><td>&lt;0.3 mmol/L</td></lln> | <0.8 - 0.6 mmol/L | <0.6 - 0.3 mmol/L | <0.3 mmol/L |
| Note: $10e9 = 10^9$ ; LLN = Lower Limit of | N = Lower Limit of N | Normal; ULN = Upper Limit of Normal | Limit of Normal | | |

Project Document Version No. Final 1.0 Project Document Effective Date: 05 April 2019 


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

Symphogen A/S Sym013-01

# 7.5 Derivation of CTCAE Grade - Coagulation Tests

| Tests | Direction | | Ğ | Grade | |
|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 |
| Activated partial | ↓ | >ULN - 1.5 x ULN >1.5 - 2.5 x ULN >2.5 x ULN; | >1.5 - 2.5 x ULN | >2.5 x ULN; | 1 |
| thromboplastin time | | | | hemorrhage | |
| prolonged | | | | | |
| Fibrinogen | <b>↑</b> | <1.0 - 0.75 x LLN | <1.0 - 0.75 x LLN <0.75 - 0.5 x LLN <0.5 - 0.25 x LLN | l | <0.25 x LLN or |
| decreased | | or <25% decrease | or $25 - <50\%$ | or $50 - < 75\%$ | 75% decrease from |
| | | from baseline | decrease from | decrease from | baseline or absolute |
| | | | baseline | baseline | value <50 mg/dL |

CONFIDENTIAL Project Document Version No. Final 1.0

Project Document Effective Date: 05 April 2019


Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

TP-GDO-WW-133-01

| Symph | ogen | A/S |
|-------|------|-----|
|-------|------|-----|

| Sym013-01 Symphogen A/S | |
|---|---|
| Sym013-01 | |
| An Open-label, Multicenter, Phase 1a/2a Trial Investigatin<br>Antitumor Activity of Multiple Doses of Sym013 (Pan-HER)<br>Targeting EGFR, HER2 and HER3, in Patients with Adva<br>Statistical Analysis Plan | , a Monoclonal Antibody Mixture |
| Symphogen A/S SIGNATURE PAGE | |
| Approved by: | |
| Li Di | April 5, 2019 |
| Cliff L. Ding, Ph.D. | Date (DD Mmm YY) |
| Statistical Consultant, Symphogen A/S | |


Page 3 of 6

Ph.D.

Date (DD)

Onsultant, Symphogen A/S

Date (DD

gis

t, Symphogen A/S

# **PAREXEL International Electronic Signature Page**

This page is the manifestation of the electronic signature(s) used in compliance with PAREXEL International's electronic signature policies and procedures and in compliance with applicable regulations.

UserName: Mattana, Flavia (mattanf) Title: Senior Biostatistician, GDO

Date: Friday, 12 April 2019, 07:52 PM GMT Standard Time

Meaning: Document contents approved.